# The incidence of venous thromboembolism in atopic dermatitis: A matched cohort analysis in UK primary care: Statistical Analysis Plan and Protocol

| <b>Document version</b> | 1.1 |
|-------------------------|-------------|
| Date | 5 July 2021 |

## Contents

| List of abbreviations | 4 |
|---------------------------------------------------------------|----|
| 1. Introduction | 5 |
| 1.1 Background | 5 |
| Atopic dermatitis | 5 |
| Venous thromboembolism | 5 |
| 1.2. Purposes of analyses | 6 |
| 2. Study objectives and endpoints | 6 |
| 2.1 Study objectives | 6 |
| 2.2 Primary objective | 6 |
| 2.3 Secondary objectives: | 6 |
| 2.4 Primary endpoint | 6 |
| 2.5 Secondary endpoints | 7 |
| 2.6 Other exploratory analyses | 7 |
| 3 General Study Design and Plan | 7 |
| 3.1 Study Design | 7 |
| 3.2 Data source and Read codes | 7 |
| 3.3 Data extraction | 7 |
| 3.4 Inclusion-Exclusion Criteria and General Study Population | 8 |
| Definition of atopic dermatitis | 8 |
| Definition of AD cases (active atopic dermatitis) | 8 |
| Definition of atopic dermatitis severity | 9 |
| Definition of Allergic conditions | 9 |
| Definition of Anticoagulant prescriptions | 9 |
| 3.5 Baseline socio-economic characteristics: | 9 |
| VTE history and established VTE risk factors | 9 |
| 4 Sample size calculations | 10 |
| 5 Populations to be analysed | 10 |

| 5.1 | Inclusion Criteria | 10 |
|----------|-----------------------------------|----|
| 5.2 | Exclusion Criteria | 10 |
| 5.3 | Matching process | 10 |
| 5.4 A | D definition exploratory analyses | 11 |
| 6 Statis | tical Analysis | 11 |
| 6.1 S | tatistical principles | 11 |
| 6.2 P | rimary Endpoint Analysis | 11 |
| 6.3 S | econdary Endpoint Analysis | 12 |
| 6.4 S | ensitivity analysis | 12 |
| 6.5 M | fissing data | 13 |
| 7 Study | Limitations | 13 |
| 8 Statis | tical software | 13 |
| 9 Ethics | S | 13 |
| Referen | nces | 15 |
| Append | dix 1 | 17 |
| Append | lix 2 | 18 |
| Append | lix 3 | 38 |
| Append | dix 4 | 45 |

# List of abbreviations

| Abbreviation | Full Form |
|---|---|
| AD | Atopic dermatitis |
| ADEPT | Anonymised Data Ethics Protocols and Transparency |
| BMI | Body mass index |
| CI | Confidence Interval |
| CKD | Chronic kidney disease |
| COPD | Chronic obstructive pulmonary disease |
| DOAC | Direct oral anticoagulant |
| DVT | Deep vein thrombosis |
| GEP | Good Epidemiological Practice |
| GP | General Practitioner |
| GPP | Good Pharmacoepidemiology Practices |
| HR | Hazard Ratio |
| HRT | Hormone replacement therapy |
| IBD | Inflammatory bowel disease |
| IEA | International Epidemiological Association |
| IMD | Index of multiple deprivation |
| IQR | Interquartile range |
| ISPE | International Society for Pharmacoepidemiology |
| OPCRD | Optimum Patient Care Research Database |
| PE | Pulmonary embolism |
| RA | Rheumatoid arthritis |
| RECORD | Reporting of studies conducted using observational routinely collected data |
| SD | Standard deviation |
| TCI | Topical calcineurin inhibitor |
| VTE | Venous thromboembolism |

## 1. Introduction

## 1.1 Background

#### Atopic dermatitis

Atopic dermatitis (AD) is a chronic inflammatory skin condition that affects around 200 million people worldwide (1). The incidence of AD has risen significantly over recent decades, in particular in high income countries (2). It most commonly develops in the first year of life, although onset can occur at any age (3, 4). AD usually follows a chronic relapsing-remitting course, and maintaining disease control may require the use of ongoing treatment (5).

Whilst many AD-affected children will have resolution or improvement by late childhood (3), a substantial proportion of people will have ongoing AD into adulthood, and flare ups can occur even after long periods of remission (4, 6). Itch, discomfort and visible skin lesions can result in disturbed sleep, social embarrassment and impaired quality of life (7).

Given that the majority of AD patients are seen and treated principally in primary care in the UK, databases of electronic health records from general practitioner (GP) practices provide a rich data source from which epidemiological analyses can be derived (8).

#### Venous thromboembolism

Venous thromboembolism (VTE), which comprises pulmonary embolism (PE) and deep vein thrombosis (DVT), is relatively common, with an incidence in the general population of around 3 cases per 1,000 patient years (9). It is associated with significant morbidity and mortality (10, 11).

VTE occurs due to a complex interplay of acquired or inherited thrombotic tendencies alongside various risk factors including active cancer, fractures, surgery, immobility, use of oral corticosteroids, superficial vein thrombosis, and in women, pregnancy and puerperium, oral contraception, and hormone therapy (12-15). In addition to these risk factors, conditions associated with chronic inflammation are increasingly being recognised as increasing the risk of VTE. Observational data demonstrate higher VTE rates in people with chronic inflammatory diseases including ulcerative colitis, Crohn's disease, rheumatoid arthritis, psoriatic arthritis, and psoriasis compared to the general population (16-21). However, to our knowledge there have not been any large population-based studies assessing the incidence of VTE in people with AD

compared to people without the condition. Studies are also lacking as to whether known risk factors carry the same risk of VTE in people with and without AD.

## 1.2. Purposes of analyses

In this retrospective population-based study we will set out to establish the presence and magnitude of any excess risk of VTE in people with AD compared to a control population without AD. We will also explore potential heterogeneity in the risk of VTE across subgroups of people with AD defined by sociodemographic factors and established VTE risk factors which are prevalent in people with AD

## 2. Study objectives and endpoints

## 2.1 Study objectives

The overall purpose of this study is to examine whether VTE is higher in people with AD compared and those without, and to explore the risk in particular subgroups of people with AD such as those with higher body mass index (BMI) or using oestrogen containing contraceptives. Such insights will be valuable for clinicians in advising patients with AD regarding VTE prevention and detection and when selecting AD treatments.

## 2.2 Primary objective

To describe the risk of VTE in people with AD compared to a matched control population.

## 2.3 Secondary objectives:

- 1) To describe the risk of PE and DVT individually in people with AD compared to a matched control population.
- 2) To explore potential heterogeneity in the risk of VTE across subgroups of people with AD: by sex, age groups (18-45, 45-65, 65+), obesity, baseline use of oestrogen containing contraceptives in females, AD severity and history of allergic conditions.

## 2.4 Primary endpoint

The primary endpoint will be a diagnosis of VTE (a composite of PE or DVT) within 10 years starting from the index date. When both PE and DVT occur, the VTE diagnosis date will be the earliest of PE or DVT.

#### 2.5 Secondary endpoints

- 1) Diagnosis of PE and diagnosis of DVT individually within 10 years starting from the index date. When both PE and DVT occur on the same event day this will be classified as a PE. Outcomes will be identified using previously validated, and subsequently updated, code lists. (22)
- 2) Diagnosis of VTE (a composite of PE or DVT) within 10 years starting from the index date.

## 2.6 Other exploratory analyses

To cover the possibility of non-recorded VTE, we will analyse a composite of VTE diagnosis in people initiated on anticoagulant prescriptions without a recorded diagnosis of atrial fibrillation or prosthetic heart value. The potential VTE event date for those without a VTE diagnosis but started on an anticoagulant will be the date of initiation of the anticoagulant.

## 3 General Study Design and Plan

## 3.1 Study Design

This is a non-interventional matched cohort study.

#### 3.2 Data source and Read codes

This study will use routinely collected and collated data from the Optimum Patient Care Research Database (OPCRD).(23) This database incorporates pseudonymised primary care records from up to 700 GP practices distributed across England, Wales, Scotland and Northern Ireland. The current OPCRD cohort size is over 5 million actively registered people, and historic records available for 10.1 million people. The cohort dataset can be enhanced through direct-to-patient and direct-to-care provider questionnaires.

#### 3.3 Data extraction

Individual patient data is anonymised at the point of data extraction. Queries will be executed to extract relevant data from the OPCRD using the Read code listed in Appendix 1. All data will remain in anonymised form and will be held on a secure server. The data will not be used for any purposes other than for the research which is described in the respective protocols and which has been approved by OPC. The sponsor, Pfizer Ltd, will not have access to the individual anonymised patient data.

## 3.4 Inclusion-Exclusion Criteria and General Study Population

#### Definition of atopic dermatitis

AD will be identified using a combination of AD specific diagnosis Read and SNOMED codes, and two or more AD treatments prescribed on different dates. Diagnosis codes which are not specific for AD (e.g., hand dermatitis) are not included for AD case finding. The full list of diagnosis codes to be used is provided in Appendix 1.

The treatments used to define AD will comprise; topical emollients, topical steroids, and topical calcineurin inhibitors. We will also make our AD case definition more stringent than that used by Abuabara et al. (24) by excluding people with conditions that may be misdiagnosed or miscoded as AD in primary care; these comprise psoriasis, contact dermatitis, photodermatitis, or ichthyosis. People with diagnosis codes for one or more of these conditions at any point in the clinical record will be excluded.

#### Definition of AD cases (active atopic dermatitis)

AD cases are defined as those people having active AD. Active AD will be identified as being present in those people prescribed one or more treatments for their AD in the last 365 days. The treatments used to define active AD comprise all those used to define AD with the addition of systemic immunomodulatory medications, including methotrexate, azathioprine, mycophenolate, cyclosporine, or AD specific biologic therapy (dupilumab being the only one licensed at during the study period). Systemic immunomodulatory medications will not be included in the AD case definition as this may lead to incorrect identification of AD cases in people with other autoimmune conditions for which these medications are used such as rheumatoid arthritis. This approach has been demonstrated to be in good agreement with physician confirmed active AD (24).

All adults with an episode of active AD at any point between 1<sup>st</sup> Jan 2010 to 1<sup>st</sup> Jan 2015 will be included for analysis. People will be eligible for inclusion as an AD case if they have a minimum of five years of possible follow up, are aged 18 and over and have AD (using an approach derived from a validated AD case definition which is described in detail elsewhere (25)) which is active at some point during the observation period.

The study period will be a ten-year period from 1<sup>st</sup> Jan 2010 to 1<sup>st</sup> Jan 2020. Individuals must enter the study on or before 1<sup>st</sup> Jan 2015 in order to have a possible minimum follow up duration

of five years. The start of follow up (index date) for each AD case will be the start of their period of active AD. Their follow-up will end at either the earliest of the following: date of deregistration, date of reaching age 95, date of death, or date of the end of the study period (1st Jan 2020).

#### Definition of atopic dermatitis severity

AD severity will be defined using the approach used by Silverwood et al. in their study of cardiovascular outcomes in AD:(26) AD will be considered moderate at the prescription of a second potent topical corticosteroid treatment within one year or a first topical calcineurin inhibitor (TCI). AD will be considered severe at the first of a systemic immunosuppressant treatment (ciclosporin, azathioprine, mycophenolate, methotrexate, and biologics), phototherapy, or a dermatology referral.

#### Definition of Allergic conditions

Allergic conditions will comprise common allergies; allergic rhinitis, allergy to dust mites or animal dander, and food allergies e.g., nut, fruit, shellfish, eggs and cows' milk allergies. Medication and other allergies will not be included.

#### Definition of Anticoagulant prescriptions

Anticoagulant prescriptions will comprise vitamin K antagonists (warfarin), low molecular weight heparins, and direct-acting oral anticoagulants.

#### 3.5 Baseline socio-economic characteristics:

Age, sex, ethnic group and socioeconomic status will comprise the sociodemographic exposures of interest. Ethnicity will be extracted from the primary care record and grouped into major UK ethnic groups; White, Black, Asian, Mixed, and Others (27). Socioeconomic status will be defined using index of multiple deprivation (IMD), the official national measure of socioeconomic status in the UK (28).

#### VTE history and established VTE risk factors

Baseline history of VTE will be extracted from the primary care record using the same definition as for the primary VTE endpoint. VTE risk factors have be selected based on existing literature demonstrating an established association with VTE (12, 19), clinical expertise, or their inclusion in the QThrombosis tool (29). These will comprise of age, BMI, smoking and alcohol use, evidence of reduced mobility, known thrombophilia, recent hospital admission (prior six months), and the presence of comorbidities; varicose vein surgery, chronic kidney disease (CKD) stages 4 or 5,

malignancy, heart failure, chronic obstructive pulmonary disease (COPD), inflammatory bowel disease (IBD) and rheumatoid arthritis (RA).

## 4 Sample size calculations

No previous studies have examined VTE risk in people with AD to provide an estimation of effect size to inform our sample size calculation. Assuming 80% power, a 1:1 ratio of AD cases to controls, and an overall probability of VTE over the study period of 1% (a conservative estimate based on a previous analysis of VTE incidence in the general population (17), a sample size of 33,899 will be required to detect a minimum clinically relevant effect size of a 20% increased risk of VTE in the AD cohort compared to population controls. We anticipate that in excess of 50,000 people in our study cohort will have an episode of active AD during the study period and so be defined as AD cases, these will be 1:1 matched to population controls providing a study cohort well in excess of this required sample size.

## 5 Populations to be analysed

#### **5.1 Inclusion Criteria**

All adult people (aged  $\geq$  18) registered with GP practices contributing data to OPCRD between January 1, 2010 and January 1, 2020, are eligible for inclusion in the study.

#### **5.2 Exclusion Criteria**

People with less than 5 years potential follow up.

People with AD that was not active during the study period.

People without AD but diagnosed with other skin conditions (psoriasis, contact dermatitis, photodermatitis, or ichthyosis).

## 5.3 Matching process

Each adult with active AD will be 1:1 matched at their index date using, nearest neighbour matching (30) to another person without AD (people never diagnosed either with AD or any exclusion skin condition (psoriasis, contact dermatitis, photodermatitis, or ichthyosis, Appendix 2) at the date of matching). Matching variables will comprise age, sex, duration of practice registration and within primary care practice where numbers allow. After matching, the index date for each control will be set at the index date of their matched counterpart.

#### 5.4 AD definition exploratory analyses

We will explore other recorded dermatology conditions to ensure that the AD case definition is correctly identifying people with AD; this analysis will be performed in practices using the Read version 2 coding system where is it possible to use search terms M1% and M2% (where % is a wild card) to extract all non-infectious dermatology diagnoses.

## **6 Statistical Analysis**

#### **6.1 Statistical principles**

The mean, standard deviation (sd) and any other statistical measures, will be reported to one decimal place. Continuous data will be summarised in the form of means, sd, median, interquartile range (IQR) and range as appropriate. Categorical data will be summarised using frequencies and proportions. Chi-squared and t-tests will be performed to compare the frequency of dichotomous variables and the values of continuous variables where relevant. 95% CIs will be reported for main effect sizes. Statistical significance will be assessed using p<0.05. Actual p-values will be reported except for p-values less than 3 decimal places which will be reported as "<0.001". P-values >0.1 will be reported to one decimal place, p-values between 0.01 and 0.1 will be reported to 2 decimal places, and p-values between 0.001 and 0.01 will be reported to three decimal places.

The assessment of any associations with baseline characteristics and the primary endpoint will be assessed using Cox proportional hazards models. A standard set of features will be used in all multivariable models as listed in section 6.2.

Assumptions of statistical approaches will be assessed, and transformations used if necessary (although it is not anticipated that the data will violate model assumptions).

## **6.2 Primary Endpoint Analysis**

Risk of new onset VTE will be assessed prospectively in AD cases and matched controls from the index date. The clinical codes used to define the VTE end points are listed in Appendix 3. Risk of developing each VTE condition within 10 years will then be examined using time to event analysis. Initially, unadjusted Cox proportional hazards models, stratified by matched set (AD cases versus matched controls), will be used to provide overall hazard ratios (HRs) as summary estimates for the association of the presence of active AD with the time to each VTE condition. Models will be

adjusted for baseline sociodemographic and clinical features, and VTE risk factors in multivariable analysis. These comprise of age, ethnicity, SES, number of primary care visits in the preceding year. BMI, smoking and alcohol use, evidence of reduced mobility, known thrombophilia, recent hospital admission (prior six months), and the presence of comorbidities; varicose vein surgery, CKD stages 4 or 5, malignancy, heart failure, COPD, IBD and RA. We will also control for active prescribing at baseline of the following medications: oral corticosteroids (which can be used in AD treatment), hormone therapy (oestrogen containing oral hormonal contraceptives, and hormone replacement therapy [HRT]), antiplatelet agents (aspirin or adenosine diphosphate receptor inhibitors), warfarin, and direct oral anticoagulants (DOACs). Hormonal contraceptives comprised only combined oestrogen and progestogen preparations; progesterone only contraceptives will not be included as these preparations are not associated with VTE (31). HRT comprises of systemic oestrogen only preparations. Active prescribing at baseline will be defined as an issued prescription in the 3 months preceding and/or 1 month after the person's start date. A full list of the study variables in included in Appendix 4.

## **6.3 Secondary Endpoint Analysis**

The secondary endpoint analysis will be assessed using the same statistical principles as the primary endpoint. Only risk of the composite VTE endpoint will be applied for the subgroup analysis.

## **6.4 Sensitivity analysis**

We will repeat the primary analysis excluding AD cases and controls (and their corresponding matched pair) with a history of VTE at cohort entry.

To evaluate the magnitude of potential bias from including as controls people who are registered with GP practices but who do not attend their practice, we will repeat the primary outcome analysis including only controls with a least one primary care consultation in the year before index date (NB this is a likely over-adjustment as the remaining controls with be less a healthy group than the general population).

To mitigate the possibility of misclassification of AD severity caused by the use of systemic treatments for other inflammatory conditions we will repeat the primary analysis and AD severity subgroup analyses in a subgroup of people without the following conditions; IBD (both ulcerative colitis and Crohn's disease) and RA.

## 6.5 Missing data

This study will use the missing indicator variable method as missing data are considered likely not to be missing at random, meaning multiple imputation approaches will lack validity.

Patients will need to be excluded from analyses based on a matched design if they have incomplete data in the fields (age, sex) required to run the matching process. In similar studies, the exclusion rate due to incomplete data has been low (32, 33).

## 7 Study Limitations

Although the data is derived from a validated and nationally representative sample of the UK, results should not be extrapolated to dissimilar populations. Important limitations of the study include the reliance on comprehensive code lists to identify any given baseline or outcome variable. This limitation is common to all studies using routinely recorded data and will be mitigated through the use of a validated approach for defining baseline and outcome parameters. (34).

Limitations exist in the amount of clinical detail presently recorded in routine primary care electronic health records. Routine primary care databases offer the benefit of large cohorts at the expense of granularity; a limitation that is universal in epidemiological studies of this type. Some analyses will be restricted to people in whom complete information is available which may introduce selection bias as a result. Finally, the data presented will be observational in nature and although attempts will be made to reduce confounding by statistical adjustment where relevant, it is not possible to exclude the possibility of residual confounding as part of the explanation for any findings.

## 8 Statistical software

All statistical analyses will be performed using R software version 3.4.1.

## 9 Ethics

This study requires approval by the Anonymised Data Ethics Protocols and Transparency (ADEPT) Committee. It has been uploaded to ClinicalTrials.gov.

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value, and rigor and follow generally accepted research practices described in Guidelines for Good Pharmacoepidemiology Practices (GPP) issued by the International Society for Pharmacoepidemiology (ISPE), and Good Epidemiological Practice (GEP) guidelines issued by the International Epidemiological Association (IEA). Study reporting will be conducted in accordance with the RECORD (Reporting of studies conducted using observational routinely collected data) guidelines (35).

#### **References**

- 1. Langan SM, Irvine AD, Weidinger S. Atopic dermatitis. The Lancet. 2020;396(10247):345-60.
- 2. Nutten S. Atopic Dermatitis: Global epidemiology and risk factors. Annal Nutri Metab. 2015;66:8-16.
- 3. Illi S, von Mutius E, Lau S, Nickel R, Gruber C, Niggemann B, et al. The natural course of atopic dermatitis from birth to age 7 years and the association with asthma. The Journal of allergy and clinical immunology. 2004;113(5):925-31.
- 4. Garmhausen D, Hagemann T, Bieber T, Dimitriou I, Fimmers R, Diepgen T, et al. Characterization of different courses of atopic dermatitis in adolescent and adult patients. Allergy. 2013;68(4):498-506.
- 5. Weidinger S, Novak N. Atopic dermatitis. Lancet (London, England). 2016;387(10023):1109-22.
- 6. Peters AS, Kellberger J, Vogelberg C, Dressel H, Windstetter D, Weinmayr G, et al. Prediction of the incidence, recurrence, and persistence of atopic dermatitis in adolescence: a prospective cohort study. The Journal of allergy and clinical immunology. 2010;126(3):590-5.e1-3.
- 7. Drucker AM, Wang AR, Li WQ, Sevetson E, Block JK, Qureshi AA. The Burden of Atopic Dermatitis: Summary of a Report for the National Eczema Association. J Invest Dermatol. 2017;137(1):26-30.
- 8. Emerson RM, Williams HC, Allen BR. Severity distribution of atopic dermatitis in the community and its relationship to secondary referral. The British journal of dermatology. 1998;139(1):73-6.
- 9. Walker AJ, Card TR, West J, Crooks C, Grainge MJ. Incidence of venous thromboembolism in patients with cancer a cohort study using linked United Kingdom databases. European journal of cancer (Oxford, England: 1990). 2013;49(6):1404-13.
- 10. Cohen AT, Agnelli G, Anderson FA, Arcelus JI, Bergqvist D, Brecht JG, et al. Venous thromboembolism (VTE) in Europe. The number of VTE events and associated morbidity and mortality. Thrombosis and haemostasis. 2007;98(4):756-64.
- 11. Winter MP, Schernthaner GH, Lang IM. Chronic complications of venous thromboembolism. Journal of thrombosis and haemostasis: JTH. 2017;15(8):1531-40.
- 12. Huerta C, Johansson S, Wallander M, García Rodríguez LA. Risk factors and short-term mortality of venous thromboembolism diagnosed in the primary care setting in the united kingdom. Archives of Internal Medicine. 2007;167(9):935-43.
- 13. Dregan A, Charlton J, Chowienczyk P, Gulliford MC. Chronic Inflammatory Disorders and Risk of Type 2 Diabetes Mellitus, Coronary Heart Disease, and Stroke. Circulation. 2014;130(10):837-44.
- 14. Zakai NA, Wright J, Cushman M. Risk factors for venous thrombosis in medical inpatients: validation of a thrombosis risk score. Journal of thrombosis and haemostasis: JTH. 2004;2(12):2156-61.
- 15. Heit JA. Epidemiology of venous thromboembolism. Nat Rev Cardiol. 2015;12(8):464-74.
- 16. Branchford BR, Carpenter SL. The Role of Inflammation in Venous Thromboembolism. Frontiers in pediatrics. 2018;6:142-.
- 17. Galloway J, Barrett K, Irving P, Khavandi K, Nijher M, Nicholson R, et al. Risk of venous thromboembolism in immune-mediated inflammatory diseases: a UK matched cohort study. RMD Open. 2020;6(3).
- 18. Choi HK, Rho Y-H, Zhu Y, Cea-Soriano L, Aviña-Zubieta JA, Zhang Y. The risk of pulmonary embolism and deep vein thrombosis in rheumatoid arthritis: a UK population-based outpatient cohort study. Annals of the Rheumatic Diseases. 2013;72(7):1182-7.

- 19. Ogdie A, Kay McGill N, Shin DB, Takeshita J, Jon Love T, Noe MH, et al. Risk of venous thromboembolism in patients with psoriatic arthritis, psoriasis and rheumatoid arthritis: a general population-based cohort study. European Heart Journal. 2018;39(39):3608-14.
- 20. Grainge MJ, West J, Card TR. Venous thromboembolism during active disease and remission in inflammatory bowel disease: a cohort study. The Lancet. 2010;375(9715):657-63.
- 21. Murthy SK, Nguyen GC. Venous Thromboembolism in Inflammatory Bowel Disease: An Epidemiological Review. The American Journal Of Gastroenterology. 2011;106:713.
- 22. Lawrenson R, Todd JC, Leydon GM, Williams TJ, Farmer RD. Validation of the diagnosis of venous thromboembolism in general practice database studies. British journal of clinical pharmacology. 2000;49(6):591-6.
- 23. OPCRD OPCRD The Optimum Patient Care Research Database 2016 [Available from: <a href="http://optimumpatientcare.org/opcrd/">http://optimumpatientcare.org/opcrd/</a>.
- 24. Abuabara K, Magyari AM, Hoffstad O, Jabbar-Lopez ZK, Smeeth L, Williams HC, et al. Development and Validation of an Algorithm to Accurately Identify Atopic Eczema Patients in Primary Care Electronic Health Records from the UK. J Invest Dermatol. 2017;137(8):1655-62.
- 25. de Lusignan S, Alexander H, Broderick C, Dennis J, McGovern A, Feeney C, et al. Epidemiology and management of atopic dermatitis in England: an observational cohort study protocol. BMJ Open. 2020;10(9):e037518.
- 26. Silverwood RJ, Forbes HJ, Abuabara K, Ascott A, Schmidt M, Schmidt SAJ, et al. Severe and predominantly active atopic eczema in adulthood and long term risk of cardiovascular disease: population based cohort study. BMJ (Clinical research ed). 2018;361:k1786.
- 27. Tippu Z, Correa A, Liyanage H, Burleigh D, McGovern A, Van Vlymen J, et al. Ethnicity Recording in Primary Care Computerised Medical Record Systems: An Ontological Approach. J Innov Health Inform. 2017;23(4):920.
- 28. Department for Communities and Local Government. The English Indices of Deprivation. 2015. [Internet; cited 2019 Jun 16]. Available from: <a href="https://www.gov.uk/government/statistics/english-indices-of-deprivation-2015">https://www.gov.uk/government/statistics/english-indices-of-deprivation-2015</a>.
- 29. Hippisley-Cox J, Coupland C. Development and validation of risk prediction algorithm (QThrombosis) to estimate future risk of venous thromboembolism: prospective cohort study. BMJ. 2011;343:d4656.
- 30. Wang SV, Schneeweiss S, Rassen JA. Optimal matching ratios in drug safety surveillance. Epidemiology. 2014;25(5):772-3.
- 31. Mantha S, Karp R, Raghavan V, Terrin N, Bauer KA, Zwicker JI. Assessing the risk of venous thromboembolic events in women taking progestin-only contraception: a meta-analysis. BMJ. 2012;345(aug07 2):e4944-e.
- 32. Kumar S, de Lusignan S, McGovern A, Correa A, Hriskova M, Gatenby P, et al. Ischaemic stroke, haemorrhage, and mortality in older patients with chronic kidney disease newly started on anticoagulation for atrial fibrillation: a population based study from UK primary care. Bmj. 2018;360:k342.
- 33. Rayner LH, Mcgovern A, Sherlock J, Gatenby P, Correa A, Creagh-Brown B, et al. The impact of therapy on the risk of asthma in type 2 diabetes. Clin Respir J. 2019;13(5):299-305.
- 34. de Lusignan S, Liaw ST, Michalakidis G, Jones S. Defining datasets and creating data dictionaries for quality improvement and research in chronic disease using routinely collected data: an ontology-driven approach. Informatics in primary care. 2011;19(3):127-34.
- 35. Benchimol EI, Smeeth L, Guttmann A, Harron K, Moher D, Petersen I, et al. The REporting of studies Conducted using Observational Routinely-collected health Data (RECORD) statement. PLoS Med. 2015;12(10):e1001885.

Diagnosis codes which will be used as part of an algorithm to identify people with atopic dermatitis. The included codes lists cover the three coding systems currently in using in UK primary care; Read V2, Read CTV3, SNOMED CT.

| Read V2 Code | Code description |
|----------------|----------------------------------------|
| M12z1 | Eczema NOS |
| M111. | Atopic dermatitis/eczema |
| M112. | Infantile eczema |
| M113. | Flexural eczema |
| M114. | Allergic (intrinsic) eczema |
| Read CTV3 Code | Description |
| X505K | Eczema |
| X505M | Constitutional eczema |
| M111. | Atopic dermatitis |
| M113. | Flexural atopic dermatitis |
| M112. | Infantile eczema |
| SNOMED CT ID | Description |
| 24079001 | Atopic dermatitis |
| 402196005 | Childhood atopic dermatitis (disorder) |
| 402195009 | Infantile atopic dermatitis (disorder) |
| 402183009 | Flexural atopic dermatitis |
| 402197001 | Adult atopic dermatitis |
| 90823000 | Infantile eczema |
| 43116000 | Eczema |
| 57092006 | Flexural eczema |

Diagnosis codes which will be used to identify AD case exclusion skin conditions.

| Psoriasis | |
|----------------|---------------------------------------------|
| Read V2 Code | Code description |
| M16 | Psoriasis and similar disorders |
| M161. | Other psoriasis |
| M1610 | Psoriasis unspecified |
| M1611 | Psoriasis annularis |
| M1612 | Psoriasis circinata |
| M1613 | Psoriasis diffusa |
| M1614 | Psoriasis discoidea |
| M1615 | Psoriasis geographica |
| M1616 | Guttate psoriasis |
| M1617 | Psoriasis gyrata |
| M1618 | Psoriasis inveterata |
| M1619 | Psoriasis ostracea |
| M161A | Psoriasis palmaris |
| M161B | Psoriasis plantaris |
| M161C | Psoriasis punctata |
| M161D | Pustular psoriasis |
| M161E | Psoriasis universalis |
| M161F | Psoriasis vulgaris |
| M161G | Acrodermatitis continua |
| M161H | Erythrodermic psoriasis |
| M161J | Flexural psoriasis |
| M161z | Psoriasis NOS |
| M166. | Palmoplantar pustular psoriasis |
| M16y. | Other psoriasis and similar disorders |
| M16y0 | Scalp psoriasis |
| M16z. | Psoriasis and similar disorders NOS |
| Myu30 | [X]Other psoriasis |
| N0452 | Juvenile arthritis in psoriasis |
| Read CTV3 Code | Description |
| X506Y | Psoriasis |
| XaYOx | Pustular psoriasis |
| X506p | Generalised pustular psoriasis |
| X506q | Acute generalised pustular psoriasis |
| X506r | Generalised pustular psoriasis of pregnancy |
| X506s | Pustular psoriasis in children |
| X506t | Juvenile pustular psoriasis |
| X506u | Infantile pustular psoriasis |
| X506l | Localised pustular psoriasis |
| X506m | Palmoplantar pustular psoriasis |
| M07y0 | Acute palmoplantar pustular psoriasis |
| M161A | Psoriasis palmaris |

| M161B | Psoriasis plantaris |
|---|---|
| X506o | Lapiere type of psoriasis |
| X506v | Circinate and annular pustular psoriasis |
| M1611 | Psoriasis annularis |
| M1612 | Psoriasis circinata |
| M1612 | |
| XaNXa | Plaque psoriasis |
| M1616 | Chronic large plaque psoriasis Guttate psoriasis |
| | · |
| X506Z<br>X506a | Flexural psoriasis |
| | Unstable psoriasis |
| X506b | Erythrodermic psoriasis |
| X506i | Scalp psoriasis |
| M161. | Other psoriasis |
| M1610 | Psoriasis unspecified |
| M1613 | Psoriasis diffusa |
| M1615 | Psoriasis geographica |
| M1617 | Psoriasis gyrata |
| M1618 | Psoriasis inveterata |
| M161C | Psoriasis punctata |
| M161E | Psoriasis universalis |
| XaNXt | Psoriasis vulgaris |
| M161z | Psoriasis NOS |
| Myu30 | [X]Other psoriasis |
| SNOMED CT ID | Description |
| 0044000 | |
| 9014002 | Psoriasis (disorder) |
| 402325007 | Drug-exacerbated psoriasis (disorder) |
| 402325007<br>402329001 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) |
| 402325007<br>402329001<br>402332003 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004<br>200977004 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004<br>200977004<br>402335001 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004<br>200977004<br>402335001<br>402336000 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004<br>200977004<br>402335001<br>402336000<br>402337009 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) Familial psoriasis without affected first degree relative (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004<br>200977004<br>402335001<br>402336000<br>402337009<br>719810000 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) Familial psoriasis without affected first degree relative (disorder) X-linked intellectual disability with seizure and psoriasis syndrome (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004<br>200977004<br>402335001<br>402336000<br>402337009<br>719810000<br>238600001 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) X-linked intellectual disability with seizure and psoriasis syndrome (disorder) Flexural psoriasis (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004<br>200977004<br>402335001<br>402336000<br>402337009<br>719810000<br>238600001<br>402317005 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) X-linked intellectual disability with seizure and psoriasis syndrome (disorder) Flexural psoriasis (disorder) Generalized psoriasis (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>4023330006<br>238603004<br>200977004<br>402335001<br>402337009<br>719810000<br>238600001<br>402317005<br>37042000 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) X-linked intellectual disability with seizure and psoriasis syndrome (disorder) Flexural psoriasis (disorder) Generalized psoriasis (disorder) Guttate psoriasis (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004<br>200977004<br>402335001<br>402336000<br>402337009<br>719810000<br>238600001<br>402317005<br>37042000<br>402312004 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) Familial psoriasis without affected first degree relative (disorder) X-linked intellectual disability with seizure and psoriasis syndrome (disorder) Flexural psoriasis (disorder) Generalized psoriasis (disorder) Guttate psoriasis (disorder) Acute guttate psoriasis (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>4023330006<br>238603004<br>200977004<br>402335001<br>402336000<br>402337009<br>719810000<br>238600001<br>402317005<br>37042000<br>402313009 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) Familial psoriasis without affected first degree relative (disorder) X-linked intellectual disability with seizure and psoriasis syndrome (disorder) Flexural psoriasis (disorder) Generalized psoriasis (disorder) Guttate psoriasis (disorder) Acute guttate psoriasis (disorder) Guttate flare of psoriasis with preexisting plaques (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004<br>200977004<br>402335001<br>402336000<br>402337009<br>719810000<br>238600001<br>402317005<br>37042000<br>402312004<br>402313009<br>402322005 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Ezzematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) X-linked intellectual disability with seizure and psoriasis syndrome (disorder) Flexural psoriasis (disorder) Generalized psoriasis (disorder) Guttate psoriasis (disorder) Acute guttate psoriasis (disorder) Guttate flare of psoriasis with preexisting plaques (disorder) Hypertrophic palmar psoriasis (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402333006<br>238603004<br>200977004<br>402335001<br>402336000<br>402337009<br>719810000<br>238600001<br>402317005<br>37042000<br>402312004<br>402313009<br>402322005<br>402323000 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) Familial psoriasis without affected first degree relative (disorder) X-linked intellectual disability with seizure and psoriasis syndrome (disorder) Flexural psoriasis (disorder) Generalized psoriasis (disorder) Guttate psoriasis (disorder) Acute guttate psoriasis (disorder) Guttate flare of psoriasis with preexisting plaques (disorder) Hypertrophic palmar psoriasis (disorder) Hypertrophic palmoplantar psoriasis (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004<br>200977004<br>402335001<br>402336000<br>402337009<br>719810000<br>238600001<br>402317005<br>37042000<br>402312004<br>402313009<br>402323000<br>238609000 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) Familial psoriasis without affected first degree relative (disorder) X-linked intellectual disability with seizure and psoriasis syndrome (disorder) Flexural psoriasis (disorder) Generalized psoriasis (disorder) Guttate psoriasis (disorder) Acute guttate psoriasis (disorder) Guttate flare of psoriasis with preexisting plaques (disorder) Hypertrophic palmoplantar psoriasis (disorder) K"bner psoriasis (disorder) |
| 402325007<br>402329001<br>402332003<br>402331005<br>402333008<br>402330006<br>238603004<br>200977004<br>402335001<br>402336000<br>402337009<br>719810000<br>238600001<br>402317005<br>37042000<br>402312004<br>402313009<br>402322005<br>402323000 | Drug-exacerbated psoriasis (disorder) Early onset psoriasis type 1 (disorder) Onset of psoriasis in adolescence (10-20 years) (disorder) Onset of psoriasis in childhood (1-10 years) (disorder) Onset of psoriasis in early adulthood (20-40 years) (disorder) Onset of psoriasis in infancy (<1 year) (disorder) Eczematized psoriasis (disorder) Erythrodermic psoriasis (disorder) Familial psoriasis with affected first degree relative (disorder) Familial psoriasis without affected first degree relative (disorder) X-linked intellectual disability with seizure and psoriasis syndrome (disorder) Flexural psoriasis (disorder) Generalized psoriasis (disorder) Guttate psoriasis (disorder) Acute guttate psoriasis (disorder) Guttate flare of psoriasis with preexisting plaques (disorder) Hypertrophic palmar psoriasis (disorder) Hypertrophic palmoplantar psoriasis (disorder) |

| 402324006 Non-pustular psoriasis of hands and feet (disorder) 402318000 Photoaggravated psoriasis (disorder) 200965009 Plaque psoriasis (disorder) 402311006 Actively extending plaque psoriasis (disorder) 402330005 Chronic small plaque psoriasis (disorder) 402330700 Chronic large plaque psoriasis (disorder) 402310007 Chronic stable plaque psoriasis (disorder) 200962007 Psoriasis annularis (disorder) 200963002 Psoriasis inclinate (disorder) 200964008 Psoriasis geographica (disorder) 200966005 Psoriasis geographica (disorder) 200966006 Psoriasis geographica (disorder) 200966007 Psoriasis of anogenital region (disorder) 402315001 Psoriasis of perianal skin (disorder) 402315002 Psoriasis of perianal skin (disorder) 402316001 Psoriasis of perianal skin (disorder) 402316002 Psoriasis of vulva (disorder) 402316003 Psoriasis of scale (disorder) 402316001 Psoriasis of scale (disorder) 402316003 Psoriasis of scale (disorder) 238606007 Psoriasi | | |
|---|---|---|
| Plaque psoriasis (disorder) 402311006 Actively extending plaque psoriasis (disorder) 402308005 Chronic small plaque psoriasis (disorder) 402309002 Chronic garge plaque psoriasis (disorder) 402307000 Chronic stable plaque psoriasis (disorder) 402310007 Chronic stable plaque psoriasis (disorder) 402310007 Psoriasis annularis (disorder) 200962007 Psoriasis annularis (disorder) 200964008 Psoriasis geographica (disorder) 200966005 Psoriasis gyrata (disorder) 200966005 Psoriasis gyrata (disorder) 200966006 Psoriasis gyrata (disorder) 200968006 Psoriasis gyrata (disorder) 200968006 Psoriasis of anogenital region (disorder) 402315002 Psoriasis of perianal skin (disorder) 402316001 Psoriasis of perianal skin (disorder) 402316001 Psoriasis of perianal skin (disorder) 402316001 Psoriasis of perianal skin (disorder) 402320002 Psoriasis of perianal skin (disorder) 402320002 Psoriasis of perianal skin (disorder) 402320002 Psoriasis of perianal skin (disorder) 402316003 Psoriasis of nall (disorder) 238606007 Psoriatic nall dystrophy (disorder) 238606007 Psoriatic nall dystrophy (disorder) 402319008 Psoriasis plantaris (disorder) 402319008 Psoriasis plantaris (disorder) 200972005 Psoriasis universalis (disorder) 200972006 Psoriasis universalis (disorder) 200973007 Psoriasis with arthropathy (disorder) 200973000 Psoriasis with arthropathy (disorder) 200973000 Psoriasis with arthropathy (disorder) 402327004 Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 402327004 Acute generalized pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis (disorder) 402326000 Juvenile pustular psoriasis (disorder) 402326000 Juvenile pustular psoriasis (disorder) 402326000 Juvenile pustular psoriasis (disorder) 402326000 Acrodermattis continua of Hallopeau (disorder) 402326000 Acrodermattis continua of Hallopeau (disorder) 402326000 Acrodermattis continua of Hallopeau (disorder) 402326000 Acropustular psoriasis of sole of foot (disorder) 402300000 Acropustular psoriasis of sole of foot (disorder) 402 | 402324006 | Non-pustular psoriasis of hands and feet (disorder) |
| 402311006 Actively extending plaque psoriasis (disorder) 402309005 Chronic small plaque psoriasis (disorder) 402307000 Chronic guttate pattern psoriasis (disorder) 402310007 Chronic stable plaque psoriasis (disorder) 402310007 Chronic stable plaque psoriasis (disorder) 200962007 Psoriasis annularis (disorder) 200963002 Psoriasis circinata (disorder) 200966005 Psoriasis gyrata (disorder) 200966005 Psoriasis gyrata (disorder) 200966005 Psoriasis gyrata (disorder) 200966006 Psoriasis of anogenital region (disorder) 402318000 Psoriasis of anogenital region (disorder) 402315001 Psoriasis of penianal skin (disorder) 402316001 Psoriasis of penianal skin (disorder) 402316001 Psoriasis of penianal skin (disorder) 402314003 Psoriasis of penianal skin (disorder) 402314003 Psoriasis of penianal skin (disorder) 402316001 Psoriasis of penianal skin (disorder) 402316001 Psoriasis of penianal skin (disorder) 402316001 Psoriasis of penianal skin (disorder) 40231002 Psoriasis of penianal skin (disorder) 402310002 Psoriasis of penianal skin (disorder) 402310003 Psoriasis of anal (disorder) 402310004 Psoriasis of penianal skin (disorder) 402310005 Psoriasis of scalp margin (disorder) 402319008 Psoriasis of scalp margin (disorder) 402319008 Psoriasis plantaris (disorder) 4020972005 Psoriasis punctata (disorder) 4020972005 Psoriasis universalis (disorder) 402327004 Psoriasis vulgaris (disorder) 402327004 Psoriasis with arthropathy (disorder) 402327006 Psoriasis with arthropathy (disorder) 402327008 Circinate and annular pustular psoriasis (disorder) 402327008 Circinate and annular pustular psoriasis (disorder) 402327000 Pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis (disorder) 402326009 Psoriasis universalis pustular psoriasis (disorder) 402326000 Psoriasis universalis pustular psoriasis (disorder) 402326000 Pustular psoriasis (disorder) 402327001 Pustular psoriasis (disorder) 402326003 Pustular psoriasis (disorder) 40236000 Pustular psoriasis (disorder) 402360000 Pustular psoriasis (disorder) 402360000 | 402318000 | Photoaggravated psoriasis (disorder) |
| 402308005 Chronic small plaque psoriasis (disorder) 402309002 Chronic guttate pattern psoriasis (disorder) 402307000 Chronic large plaque psoriasis (disorder) 402310007 Chronic large plaque psoriasis (disorder) 200962007 Psoriasis annularis (disorder) 200963000 Psoriasis circinata (disorder) 200964008 Psoriasis diffusa (disorder) 200966005 Psoriasis geographica (disorder) 200968006 Psoriasis geographica (disorder) 200968006 Psoriasis inveterata (disorder) 200968006 Psoriasis of anogenital region (disorder) 402315002 Psoriasis of penis (disorder) 402315002 Psoriasis of penis (disorder) 402316001 Psoriasis of penis (disorder) 402316001 Psoriasis of penis (disorder) 40231000 Psoriasis of penis (disorder) 402320002 Psoriasis of penis (disorder) 40232000 Psoriasis of face (disorder) 238604005 Psoriasis of nall (disorder) 238605006 Psoriasis of indi (disorder) 238605006 Psoriasis of indi (disorder) 238605006 Psoriasis of so fall (disorder) 238605007 Psoriasis of indi (disorder) 200971003 Psoriasis of solap margin (disorder) 200972005 Psoriasis plantaris (disorder) 200972005 Psoriasis universalis (disorder) 200973000 Psoriasis universalis (disorder) 238602009 Psoriasis with arthropathy (disorder) 238602009 Psoriasis with arthropathy (disorder) 238602009 Psoriasis with arthropathy (disorder) 238602009 Psoriasis with arthropathy (disorder) 238612000 Generalized pustular psoriasis (disorder) 238612001 Generalized pustular psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 238612003 Generalized pustular psoriasis (disorder) 238612004 Infantile pustular psoriasis (disorder) 238612005 Generalized pustular psoriasis (disorder) 238612006 Lapiere type of psoriasis (disorder) 238612007 Generalized pustular psoriasis (disorder) 238612009 Psoriasis of palma and soles (disorder) 238612000 Juvenile pustular psoriasis (disorder) 238612000 Pustular psoriasis of palma and soles (disorder) 238612000 Pustular psoriasis of palma and soles (disorder) 238612001 Pustular psoriasis of palma and soles (disorder) 23809800 | 200965009 | Plaque psoriasis (disorder) |
| 402307000 Chronic guttate pattern psoriasis (disorder) 402310007 Chronic large plaque psoriasis (disorder) 402310007 Chronic stable plaque psoriasis (disorder) 200962007 Psoriasis annularis (disorder) 200964008 Psoriasis diffusa (disorder) 200966005 Psoriasis gegraphica (disorder) 200967001 Psoriasis gyrata (disorder) 200967001 Psoriasis gyrata (disorder) 200968006 Psoriasis inveterata (disorder) 200968006 Psoriasis inveterata (disorder) 200968006 Psoriasis inveterata (disorder) 200968006 Psoriasis of penis (disorder) 200968006 Psoriasis of penis (disorder) 200968000 Psoriasis of penis (disorder) 20031000 Psoriasis of penis (disorder) 402315001 Psoriasis of penis (disorder) 402316001 Psoriasis of face (disorder) 402316003 Psoriasis of face (disorder) 402320002 Psoriasis of face (disorder) 238604005 Psoriasis of intil (disorder) 238606006 Psoriatic nail dystrophy (disorder) 238606007 Psoriasis of scalp margin (disorder) 402319008 Psoriasis of scalp margin (disorder) 200971003 Psoriasis punctata (disorder) 200972005 Psoriasis punctata (disorder) 200975007 Psoriasis universalis (disorder) 238602009 Psoriasis universalis (disorder) 238602009 Psoriasis universalis (disorder) 238602009 Psoriasis universalis (disorder) 238602009 Psoriasis wildaris (disorder) 238612004 Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 238612004 Generalized pustular psoriasis (disorder) 238612005 Generalized pustular psoriasis (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Generalized pustular psoriasis (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Pustular psoriasis (disorder) 23861000 Pustular psoriasis (disorder) 23861000 Pustular psori | 402311006 | Actively extending plaque psoriasis (disorder) |
| 402307000 Chronic large plaque psoriasis (disorder) 402310007 Chronic stable plaque psoriasis (disorder) 200962007 Psoriasis annularis (disorder) 200964008 Psoriasis circinata (disorder) 200964008 Psoriasis circinata (disorder) 200966005 Psoriasis geographica (disorder) 200966006 Psoriasis geographica (disorder) 200968006 Psoriasis geographica (disorder) 200968006 Psoriasis inveterata (disorder) 201968006 Psoriasis inveterata (disorder) 201988000 Psoriasis of anogenital region (disorder) 402315002 Psoriasis of penis (disorder) 402315001 Psoriasis of penis (disorder) 402316001 Psoriasis of penis (disorder) 402314003 Psoriasis of face (disorder) 402314003 Psoriasis of face (disorder) 402320002 Psoriasis of face (disorder) 2038604005 Psoriatic nall dystrophy (disorder) 238606006 Psoriatic nall dystrophy (disorder) 238606007 Psoriasis plantaris (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis plantaris (disorder) 200972005 Psoriasis universalis (disorder) 200975007 Psoriasis vulgaris (disorder) 23860209 Psoriasis vulgaris (disorder) 23860209 Psoriasis vulgaris (disorder) 238602009 Psoriasis ezerma overlap condition (disorder) 200973000 Pustular psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 238612003 Acute generalized pustular psoriasis (disorder) 238613007 Generalized pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 238616004 Infantile pustular psoriasis (disorder) 238616004 Infantile pustular psoriasis (disorder) 238616004 Lapiere type of psoriasis (disorder) 238616004 Lapiere type of psoriasis (disorder) 238616004 Psoriasis of palma and soles (disorder) 238616005 Psoriasis of palma and soles | 402308005 | Chronic small plaque psoriasis (disorder) |
| 402310007 Chronic stable plaque psoriasis (disorder) 200962007 Psoriasis annularis (disorder) 200964008 Psoriasis circinata (disorder) 200964008 Psoriasis geographica (disorder) 200967001 Psoriasis geographica (disorder) 200967001 Psoriasis gyrata (disorder) 200968006 Psoriasis inveterata (disorder) 200968006 Psoriasis of anogenital region (disorder) 200968006 Psoriasis of penis (disorder) 201938000 Psoriasis of penis (disorder) 402315002 Psoriasis of penis (disorder) 402315001 Psoriasis of penis (disorder) 402314003 Psoriasis of penis (disorder) 402314003 Psoriasis of face (disorder) 402320002 Psoriasis of face (disorder) 238604005 Psoriasis of face (disorder) 238605006 Psoriatic nail dystrophy (disorder) 238606007 Psoriasis of nail (disorder) 238606007 Psoriasis of scalp margin (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis plantaris (disorder) 200974006 Psoriasis plantaris (disorder) 200975007 Psoriasis vulyaris (disorder) 238602009 Psoriasis vulyaris (disorder) 238602009 Psoriasis vulyaris (disorder) 402327004 Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 402327004 Acute generalized pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis (disorder) 238612000 Generalized pustular psoriasis (disorder) 238613007 Generalized pustular psoriasis (disorder) 238613007 Generalized pustular psoriasis (disorder) 238613000 Juvenile pustular psoriasis (disorder) 238613000 Juvenile pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 238613000 Generalized pustular psoriasis (disorder) 238613000 Juvenile pustular psoriasis (disorder) 238613000 Juvenile pustular psoriasis (disorder) 238613000 Juvenile pustular psoriasis (disorder) 238613000 Pustular psoriasis (disorder) 238613000 Juvenile pustular psoriasis (disorder) 238613000 Pustular psoriasis (disorder) 238613000 Pustular psoriasis (disorder) 238613000 Pustular psoriasis of palm of hand (disorder) 238613000 Pustular psoriasis of palm of hand (disorder) 23809000 Acropus | 402309002 | Chronic guttate pattern psoriasis (disorder) |
| 200962007 Psoriasis annularis (disorder) 200964008 Psoriasis diffusa (disorder) 200966005 Psoriasis gegraphica (disorder) 200967001 Psoriasis gyrata (disorder) 200968006 Psoriasis gyrata (disorder) 200968000 Psoriasis of panis (disorder) 402315002 Psoriasis of penis (disorder) 402316001 Psoriasis of penis (disorder) 402314003 Psoriasis of penial skin (disorder) 402320002 Psoriasis of face (disorder) 238604005 Psoriasis of nail (disorder) 238605006 Psoriatic nail dystrophy (disorder) 238606007 Psoriatic nail dystrophy (disorder) 200971003 Psoriasis of scalp margin (disorder) 200972005 Psoriasis plantaris (disorder) 200972005 Psoriasis plantaris (disorder) 200975007 Psoriasis universalis (disorder) 200975007 Psoriasis with arthropathy (disorder) 238602009 Psoriasis with arthropathy (disorder) 238602009 Psoriasis with arthropathy (disorder) 238617008 Circinate and annular pustular psoriasis (disorder) <t< td=""><td>402307000</td><td>Chronic large plaque psoriasis (disorder)</td></t<> | 402307000 | Chronic large plaque psoriasis (disorder) |
| 200963002 Psoriasis circinata (disorder) 200964008 Psoriasis geographica (disorder) 200967001 Psoriasis gyrata (disorder) 200967001 Psoriasis gyrata (disorder) 200967001 Psoriasis gyrata (disorder) 200968006 Psoriasis of sonogenital region (disorder) 402315002 Psoriasis of penias (disorder) 402315001 Psoriasis of penianal skin (disorder) 402314003 Psoriasis of penianal skin (disorder) 402320002 Psoriasis of face (disorder) 238604005 Psoriasis of face (disorder) 238605006 Psoriasis of nail (disorder) 238605007 Psoriasis of scalp margin (disorder) 402319008 Psoriasis plantaris (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis punctata (disorder) 200974006 Psoriasis vulgaris (disorder) 200975007 Psoriasis with arthropathy (disorder) 23860209 Psoriasis with arthropathy (disorder) 238612009 Psoriasis with arthropathy (disorder) 238612009 Psoriasis valuar psoriasis (disorder) 23861 | 402310007 | Chronic stable plaque psoriasis (disorder) |
| 200964008 Psoriasis diffusa (disorder) 200966005 Psoriasis geographica (disorder) 200968006 Psoriasis gryrata (disorder) 200968006 Psoriasis prata (disorder) 200968000 Psoriasis of anogenital region (disorder) 402315002 Psoriasis of penis (disorder) 402316001 Psoriasis of penis (disorder) 402314003 Psoriasis of face (disorder) 238604005 Psoriasis of face (disorder) 238605006 Psoriasis of nail (disorder) 238606007 Psoriatic nail dystrophy (disorder) 238606007 Psoriatic nail pitting (disorder) 200971003 Psoriasis of scalp margin (disorder) 200972005 Psoriasis punctata (disorder) 200974006 Psoriasis universalis (disorder) 200975007 Psoriasis universalis (disorder) 238602009 Psoriasis with arthropathy (disorder) 238602009 Psoriasis with arthropathy (disorder) 238617008 Circinate and annular pustular psoriasis (disorder) 238617008 Circinate and annular pustular psoriasis (disorder) 238613007 Generalized pustular psoriasis (disorder) | 200962007 | Psoriasis annularis (disorder) |
| Psoriasis geographica (disorder) | 200963002 | Psoriasis circinata (disorder) |
| 200967001 Psoriasis gyrata (disorder) 200968006 Psoriasis inveterata (disorder) 721538000 Psoriasis of anogenital region (disorder) 402315002 Psoriasis of penis (disorder) 402316001 Psoriasis of perianal skin (disorder) 402314003 Psoriasis of vulva (disorder) 402320002 Psoriasis of face (disorder) 238604005 Psoriasis of nail (disorder) 238605006 Psoriatic nail dystrophy (disorder) 238606007 Psoriasis of scalp margin (disorder) 402319008 Psoriasis plantaris (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis plantaris (disorder) 200974006 Psoriasis vulgaris (disorder) 200975007 Psoriasis with arthropathy (disorder) 200973000 Psoriasis vulgaris (disorder) 200973000 Psoriasis vulgaris (disorder) 402327004 Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 238612002 Generalized pustular psoriasis of pregnancy (disorder) 238613007 Generalized | 200964008 | Psoriasis diffusa (disorder) |
| 200968006 Psoriasis inveterata (disorder) 721538000 Psoriasis of anogenital region (disorder) 402315002 Psoriasis of penis (disorder) 402316001 Psoriasis of perianal skin (disorder) 402314003 Psoriasis of vulva (disorder) 402320002 Psoriasis of face (disorder) 238604005 Psoriasis of nail (disorder) 238605006 Psoriatic nail dystrophy (disorder) 238606007 Psoriasis of scalp margin (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis punctata (disorder) 200974006 Psoriasis universalis (disorder) 200975007 Psoriasis with arthropathy (disorder) 238602009 Psoriasis with arthropathy (disorder) 200973000 Pustular psoriasis (disorder) 200973000 Pustular psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 238613007 Generalized pustular psoriasis (disorder) 238613007 Generalized pustular psoriasis (disorder) 238613007 Generalized pustular psoriasis (dis | 200966005 | Psoriasis geographica (disorder) |
| Psoriasis of anogenital region (disorder) 402315002 Psoriasis of penis (disorder) 402316001 Psoriasis of penis (disorder) 402314003 Psoriasis of perianal skin (disorder) 402314003 Psoriasis of fulva (disorder) 402320002 Psoriasis of face (disorder) 238604005 Psoriasis of nail (disorder) 238605006 Psoriatic nail dystrophy (disorder) 238606007 Psoriatic nail pitting (disorder) 402319008 Psoriasis of scalp margin (disorder) 402319008 Psoriasis plantaris (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis punctata (disorder) 200975007 Psoriasis universalis (disorder) 200975007 Psoriasis vulgaris (disorder) 238602009 Psoriasis vulgaris (disorder) 238602009 Psoriasis-eczema overlap condition (disorder) 402327004 Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 402327004 Acute generalized pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis de novo (disorder) 402326008 Acute generalized pustular psoriasis de novo (disorder) 238613007 Generalized pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 238611009 Lapiere type of psoriasis (disorder) 82861009 Lapiere type of psoriasis (disorder) 828611009 Lapiere type of psoriasis (disorder) 828612000 Pustular psoriasis (disorder) 828612001 Generalized pustular psoriasis (disorder) 828612002 Pustular psoriasis (disorder) 828612003 Pustular psoriasis (disorder) 828612004 Infantile pustular psoriasis (disorder) 828612009 Lapiere type of psoriasis (disorder) 828612000 Pustular psoriasis (disorder) 828612001 Generalized pustular psoriasis (disorder) 828612002 Pustular psoriasis of palm of hand (disorder) 82862000 Pustular psoriasis of palm of hand (disorder) 82862000 Pustular psoriasis of polm of hand (disorder) 82862000 Pustular psoriasis of polm of hand (disorder) 82862000 Pustular psoriasis of polm of hand (disorder) 828000 Pustular psoriasis of polm of hand (disorder) | 200967001 | Psoriasis gyrata (disorder) |
| 402315002 Psoriasis of penis (disorder) 402316001 Psoriasis of perianal skin (disorder) 402314003 Psoriasis of vulva (disorder) 402320002 Psoriasis of nail (disorder) 238604005 Psoriasis of nail (disorder) 238605006 Psoriatic nail dystrophy (disorder) 238605006 Psoriatic nail dystrophy (disorder) 238606007 Psoriatic nail dystrophy (disorder) 402319008 Psoriasis of scalp margin (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis punctata (disorder) 200974006 Psoriasis universalis (disorder) 200975007 Psoriasis vulgaris (disorder) 233339001 Psoriasis with arthropathy (disorder) 238602009 Psoriasis eczema overlap condition (disorder) 200973000 Pustular psoriasis (disorder) 402327004 Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis de novo (disorder) 238613007 Generalized pustular psoriasis of pregnancy (disorder) 238615000 Juvenile pustular psoriasis (disorder) 238611009 Lapiere type of psoriasis (disorder) 238611009 Lapiere type of psoriasis (disorder) 238611009 Lapiere type of psoriasis (disorder) 238611009 Lapiere type of psoriasis (disorder) 23861000 Pustular psoriasis of palm of hand (disorder) 238000 Pustular psoriasis of palm of hand (disorder) 2422001 Pustular psoriasis of palm of hand (disorder) 2422000 Pustular psoriasis of palm of hand (disorder) 2422000 Pustular psoriasis of palm of hand (disorder) 24222000 Pustular psoriasis of palm of hand (disorder) 24222000 Pustular psoriasis of palm of hand (disorder) 24222000 Pustular psoriasis of palm of hand (disorder) 24222000 Pustular psoriasis of palm of hand (disorder) | 200968006 | Psoriasis inveterata (disorder) |
| 402316001 Psoriasis of perianal skin (disorder) | 721538000 | Psoriasis of anogenital region (disorder) |
| 402314003 Psoriasis of vulva (disorder) 402320002 Psoriasis of face (disorder) 238604005 Psoriasis of nail (disorder) 238605006 Psoriatic nail dystrophy (disorder) 238606007 Psoriatic nail pitting (disorder) 40231908 Psoriasis of scalp margin (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis punctata (disorder) 200974006 Psoriasis universalis (disorder) 200975007 Psoriasis vulgaris (disorder) 200975007 Psoriasis with arthropathy (disorder) 238602009 Psoriasis-eczema overlap condition (disorder) 200973000 Pustular psoriasis (disorder) 402327004 Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis (disorder) 238613007 Generalized pustular psoriasis of pregnancy (disorder) 238616004 Infantile pustular psoriasis (disorder) 23861009 Lapiere type of psoriasis (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Psoriasis of pregnancy (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Psoriasis of pregnancy (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Psoriasis of psoriasis (disorder) 23861000 Psoriasis of psoriasis (disorder) 23861000 Psoriasis of psoriasis (disorder) 23861000 Psoriasis of psoriasis (disorder) 23861000 Psoriasis of palm of hand (disorder) 23861000 Pustular psoriasis of palms and soles (disorder) 238000 Psoriasis of palms and soles (disorder) 239098009 Acropustulosis of infancy (disorder) 24322005 Psutular psoriasis of sole of foot (disorder) | 402315002 | |
| 402320002 Psoriasis of face (disorder) 238604005 Psoriasis of nail (disorder) 238605006 Psoriatic nail dystrophy (disorder) 238606007 Psoriatic nail pitting (disorder) 402319008 Psoriasis of scalp margin (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis punctata (disorder) 200974006 Psoriasis universalis (disorder) 200975007 Psoriasis vulgaris (disorder) 200975007 Psoriasis vulgaris (disorder) 238602009 Psoriasis-eczema overlap condition (disorder) 200973000 Pustular psoriasis (disorder) 200973000 Pustular psoriasis (disorder) 238617008 Circinate and annular pustular psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 238613007 Generalized pustular psoriasis of pregnancy (disorder) 238613007 Generalized pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 23861004 Infantile pustular psoriasis (disorder) 23861009 Lapiere type of psoriasis (disorder) 23861000 Lapiere type of psoriasis (disorder) 23861000 Pustular psoriasis of palm of hand (disorder) 238000 Pustular psoriasis of palms and soles (disorder) 24328000 Pustular psoriasis of palms and soles (disorder) 24328000 Pustular psoriasis of sole of foot (disorder) 24327005 Pustular psoriasis of sole of foot (disorder) | 402316001 | Psoriasis of perianal skin (disorder) |
| 238604005 Psoriasis of nail (disorder) 238605006 Psoriatic nail dystrophy (disorder) 238606007 Psoriatic nail pitting (disorder) 402319008 Psoriasis of scalp margin (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis punctata (disorder) 200974006 Psoriasis universalis (disorder) 200975007 Psoriasis vulgaris (disorder) 23339001 Psoriasis with arthropathy (disorder) 238602009 Psoriasis-eczema overlap condition (disorder) 200973000 Pustular psoriasis (disorder) 238617008 Circinate and annular pustular psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 238613007 Generalized pustular psoriasis de novo (disorder) 238613007 Generalized pustular psoriasis (disorder) 238616004 Infantile pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 23861000 Generalized pustular psoriasis (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Pustular psoriasis (disorder) 23861000 Pustular psoriasis (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Pustular psoriasis of palm of hand (disorder) 24322001 Pustular psoriasis of palms and soles (disorder) 24322001 Pustular psoriasis of palms and soles (disorder) 24322001 Pustular psoriasis of sole of foot (disorder) 24322005 Pustular psoriasis (disorder) | 402314003 | Psoriasis of vulva (disorder) |
| 238605006 Psoriatic nail dystrophy (disorder) 238606007 Psoriatic nail pitting (disorder) 402319008 Psoriasis of scalp margin (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis punctata (disorder) 200974006 Psoriasis universalis (disorder) 200975007 Psoriasis vulgaris (disorder) 23339901 Psoriasis with arthropathy (disorder) 238602009 Psoriasis-eczema overlap condition (disorder) 200973000 Pustular psoriasis (disorder) 402327004 Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis (disorder) 238613007 Generalized pustular psoriasis of pregnancy (disorder) 238616004 Infantile pustular psoriasis (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Generalized pustular psoriasis (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Pustular psoriasis (disorder) 23861000 Pustular psoriasis (disorder) 23861000 Juvenile pustular psoriasis (disorder) 23861000 Pustular psoriasis (disorder) 23861000 Lapiere type of psoriasis (disorder) 23861000 Pustular psoriasis (disorder) 23861000 Pustular psoriasis (disorder) 23861000 Pustular psoriasis (disorder) 23861000 Pustular psoriasis (disorder) 23861000 Pustular psoriasis of palm of hand (disorder) 24328000 Pustular psoriasis of palms and soles (disorder) 24328000 Pustular psoriasis of palms and soles (disorder) 24327005 Pustular psoriasis of sole of foot (disorder) | 402320002 | Psoriasis of face (disorder) |
| 238606007 Psoriatic nail pitting (disorder) 402319008 Psoriasis of scalp margin (disorder) 200971003 Psoriasis plantaris (disorder) 200972005 Psoriasis punctata (disorder) 200974006 Psoriasis universalis (disorder) 200975007 Psoriasis vulgaris (disorder) 23339001 Psoriasis with arthropathy (disorder) 238602009 Psoriasis-eczema overlap condition (disorder) 200973000 Pustular psoriasis (disorder) 402327004 Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 238617008 Circinate and annular pustular psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis de novo (disorder) 238613007 Generalized pustular psoriasis of pregnancy (disorder) 238615000 Juvenile pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 23861009 Lapiere type of psoriasis (disorder) 81271001 Localized pustular psoriasis (disorder) 83839005 Acrodermatitis continua of Hallopeau (disorder) 784328000 Pustular psoriasis of palm of hand (disorder) 239098009 Acropustulosis of infancy (disorder) 230998009 Rupioid psoriasis of sole of foot (disorder) | 238604005 | Psoriasis of nail (disorder) |
| 402319008Psoriasis of scalp margin (disorder)200971003Psoriasis plantaris (disorder)200972005Psoriasis punctata (disorder)200974006Psoriasis universalis (disorder)200975007Psoriasis vulgaris (disorder)33339001Psoriasis with arthropathy (disorder)238602009Psoriasis-eczema overlap condition (disorder)200973000Pustular psoriasis (disorder)402327004Acute generalized pustular flare of preexisting plaque psoriasis (disorder)238612002Generalized pustular psoriasis (disorder)402326008Acute generalized pustular psoriasis (disorder)238613007Generalized pustular psoriasis of pregnancy (disorder)238616004Infantile pustular psoriasis (disorder)238615000Juvenile pustular psoriasis (disorder)28840001Generalized pustular psoriasis (disorder)238611009Lapiere type of psoriasis (disorder)81271001Localized pustular psoriasis (disorder)83839005Acrodermatitis continua of Hallopeau (disorder)784328000Pustular psoriasis of palm of hand (disorder)27520001Pustular psoriasis of palms and soles (disorder)239098009Acropustulosis of infancy (disorder)200969003Rupioid psoriasis (disorder) | 238605006 | Psoriatic nail dystrophy (disorder) |
| 200971003Psoriasis plantaris (disorder)200972005Psoriasis punctata (disorder)200974006Psoriasis universalis (disorder)200975007Psoriasis vulgaris (disorder)33339001Psoriasis with arthropathy (disorder)238602009Psoriasis-eczema overlap condition (disorder)200973000Pustular psoriasis (disorder)402327004Acute generalized pustular flare of preexisting plaque psoriasis (disorder)238612002Generalized pustular psoriasis (disorder)402326008Acute generalized pustular psoriasis (disorder)238613007Generalized pustular psoriasis of pregnancy (disorder)238616004Infantile pustular psoriasis (disorder)238615000Juvenile pustular psoriasis (disorder)28840001Generalized pustular psoriasis (disorder)238611009Lapiere type of psoriasis (disorder)81271001Localized pustular psoriasis (disorder)83839005Acrodermatitis continua of Hallopeau (disorder)784328000Pustular psoriasis of palms and soles (disorder)27520001Pustular psoriasis of sole of foot (disorder)23909809Acropustulosis of infancy (disorder)84327005Pustular psoriasis (disorder)200969003Rupioid psoriasis (disorder) | 238606007 | Psoriatic nail pitting (disorder) |
| 200972005Psoriasis punctata (disorder)200974006Psoriasis universalis (disorder)200975007Psoriasis vulgaris (disorder)33339001Psoriasis with arthropathy (disorder)238602009Psoriasis-eczema overlap condition (disorder)200973000Pustular psoriasis (disorder)402327004Acute generalized pustular flare of preexisting plaque psoriasis (disorder)238617008Circinate and annular pustular psoriasis (disorder)238612002Generalized pustular psoriasis (disorder)402326008Acute generalized pustular psoriasis de novo (disorder)238613007Generalized pustular psoriasis of pregnancy (disorder)238616004Infantile pustular psoriasis (disorder)238615000Juvenile pustular psoriasis (disorder)2384001Generalized pustular psoriasis, exanthematous type (disorder)238611009Lapiere type of psoriasis (disorder)81271001Localized pustular psoriasis (disorder)83839005Acrodermatitis continua of Hallopeau (disorder)784328000Pustular psoriasis of palm of hand (disorder)27520001Pustular psoriasis of palms and soles (disorder)239098009Acropustulosis of infancy (disorder)784327005Pustular psoriasis of sole of foot (disorder)200969003Rupioid psoriasis (disorder) | 402319008 | Psoriasis of scalp margin (disorder) |
| 200974006Psoriasis universalis (disorder)200975007Psoriasis vulgaris (disorder)33339001Psoriasis with arthropathy (disorder)238602009Psoriasis-eczema overlap condition (disorder)200973000Pustular psoriasis (disorder)402327004Acute generalized pustular flare of preexisting plaque psoriasis (disorder)238617008Circinate and annular pustular psoriasis (disorder)238612002Generalized pustular psoriasis (disorder)402326008Acute generalized pustular psoriasis de novo (disorder)238613007Generalized pustular psoriasis of pregnancy (disorder)238616004Infantile pustular psoriasis (disorder)238615000Juvenile pustular psoriasis (disorder)28840001Generalized pustular psoriasis, exanthematous type (disorder)238611009Lapiere type of psoriasis (disorder)81271001Localized pustular psoriasis (disorder)83839005Acrodermatitis continua of Hallopeau (disorder)784328000Pustular psoriasis of palm of hand (disorder)27520001Pustular psoriasis of palms and soles (disorder)239098009Acropustulosis of infancy (disorder)784327005Pustular psoriasis of sole of foot (disorder)200969003Rupioid psoriasis (disorder) | 200971003 | Psoriasis plantaris (disorder) |
| Psoriasis vulgaris (disorder) 33339001 Psoriasis with arthropathy (disorder) 238602009 Psoriasis-eczema overlap condition (disorder) 200973000 Pustular psoriasis (disorder) 402327004 Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 238617008 Circinate and annular pustular psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis de novo (disorder) 238613007 Generalized pustular psoriasis of pregnancy (disorder) 238616004 Infantile pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 28840001 Generalized pustular psoriasis, exanthematous type (disorder) 238611009 Lapiere type of psoriasis (disorder) 81271001 Localized pustular psoriasis (disorder) Acrodermatitis continua of Hallopeau (disorder) 784328000 Pustular psoriasis of palm of hand (disorder) 239098009 Acropustulosis of infancy (disorder) 84327005 Pustular psoriasis of sole of foot (disorder) Rupioid psoriasis (disorder) | 200972005 | Psoriasis punctata (disorder) |
| 33339001Psoriasis with arthropathy (disorder)238602009Psoriasis-eczema overlap condition (disorder)200973000Pustular psoriasis (disorder)402327004Acute generalized pustular flare of preexisting plaque psoriasis (disorder)238617008Circinate and annular pustular psoriasis (disorder)238612002Generalized pustular psoriasis (disorder)402326008Acute generalized pustular psoriasis de novo (disorder)238613007Generalized pustular psoriasis of pregnancy (disorder)238615000Juvenile pustular psoriasis (disorder)238615000Juvenile pustular psoriasis (disorder)238611009Lapiere type of psoriasis (disorder)81271001Localized pustular psoriasis (disorder)83839005Acrodermatitis continua of Hallopeau (disorder)784328000Pustular psoriasis of palm of hand (disorder)27520001Pustular psoriasis of palms and soles (disorder)239098009Acropustulosis of infancy (disorder)784327005Pustular psoriasis of sole of foot (disorder)200969003Rupioid psoriasis (disorder) | 200974006 | Psoriasis universalis (disorder) |
| Psoriasis-eczema overlap condition (disorder) 200973000 Pustular psoriasis (disorder) 402327004 Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 238617008 Circinate and annular pustular psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis de novo (disorder) 238613007 Generalized pustular psoriasis of pregnancy (disorder) 238616004 Infantile pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 23840001 Generalized pustular psoriasis, exanthematous type (disorder) 238611009 Lapiere type of psoriasis (disorder) 81271001 Localized pustular psoriasis (disorder) 83839005 Acrodermatitis continua of Hallopeau (disorder) 784328000 Pustular psoriasis of palm of hand (disorder) 239098009 Acropustulosis of infancy (disorder) 84327005 Pustular psoriasis of sole of foot (disorder) 8upioid psoriasis (disorder) | 200975007 | Psoriasis vulgaris (disorder) |
| 200973000Pustular psoriasis (disorder)402327004Acute generalized pustular flare of preexisting plaque psoriasis (disorder)238617008Circinate and annular pustular psoriasis (disorder)238612002Generalized pustular psoriasis (disorder)402326008Acute generalized pustular psoriasis de novo (disorder)238613007Generalized pustular psoriasis of pregnancy (disorder)238616004Infantile pustular psoriasis (disorder)238615000Juvenile pustular psoriasis (disorder)28840001Generalized pustular psoriasis, exanthematous type (disorder)238611009Lapiere type of psoriasis (disorder)81271001Localized pustular psoriasis (disorder)83839005Acrodermatitis continua of Hallopeau (disorder)784328000Pustular psoriasis of palm of hand (disorder)27520001Pustular psoriasis of palms and soles (disorder)239098009Acropustulosis of infancy (disorder)784327005Pustular psoriasis of sole of foot (disorder)200969003Rupioid psoriasis (disorder) | 33339001 | Psoriasis with arthropathy (disorder) |
| Acute generalized pustular flare of preexisting plaque psoriasis (disorder) 238617008 Circinate and annular pustular psoriasis (disorder) 238612002 Generalized pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis de novo (disorder) 238613007 Generalized pustular psoriasis of pregnancy (disorder) 238616004 Infantile pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 28840001 Generalized pustular psoriasis, exanthematous type (disorder) 238611009 Lapiere type of psoriasis (disorder) 81271001 Localized pustular psoriasis (disorder) 83839005 Acrodermatitis continua of Hallopeau (disorder) 784328000 Pustular psoriasis of palm of hand (disorder) 27520001 Pustular psoriasis of palms and soles (disorder) 239098009 Acropustulosis of infancy (disorder) Pustular psoriasis of sole of foot (disorder) Rupioid psoriasis (disorder) | 238602009 | Psoriasis-eczema overlap condition (disorder) |
| Circinate and annular pustular psoriasis (disorder) Generalized pustular psoriasis (disorder) Acute generalized pustular psoriasis de novo (disorder) Generalized pustular psoriasis de novo (disorder) Generalized pustular psoriasis of pregnancy (disorder) Infantile pustular psoriasis (disorder) Juvenile pustular psoriasis (disorder) Sesson Generalized pustular psoriasis (disorder) Ease of psoriasis (disorder) Lapiere type of psoriasis (disorder) Lapiere type of psoriasis (disorder) Localized pustular psoriasis (disorder) Acrodermatitis continua of Hallopeau (disorder) Pustular psoriasis of palm of hand (disorder) Pustular psoriasis of palms and soles (disorder) Acropustulosis of infancy (disorder) Pustular psoriasis of sole of foot (disorder) Rupioid psoriasis (disorder) | 200973000 | Pustular psoriasis (disorder) |
| 238612002 Generalized pustular psoriasis (disorder) 402326008 Acute generalized pustular psoriasis de novo (disorder) 238613007 Generalized pustular psoriasis of pregnancy (disorder) 238616004 Infantile pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 28840001 Generalized pustular psoriasis, exanthematous type (disorder) 238611009 Lapiere type of psoriasis (disorder) 81271001 Localized pustular psoriasis (disorder) 83839005 Acrodermatitis continua of Hallopeau (disorder) 784328000 Pustular psoriasis of palm of hand (disorder) 27520001 Pustular psoriasis of palms and soles (disorder) 239098009 Acropustulosis of infancy (disorder) 784327005 Pustular psoriasis of sole of foot (disorder) 200969003 Rupioid psoriasis (disorder) | 402327004 | Acute generalized pustular flare of preexisting plaque psoriasis (disorder) |
| Acute generalized pustular psoriasis de novo (disorder) 238613007 Generalized pustular psoriasis of pregnancy (disorder) 238616004 Infantile pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 28840001 Generalized pustular psoriasis, exanthematous type (disorder) 238611009 Lapiere type of psoriasis (disorder) 81271001 Localized pustular psoriasis (disorder) 83839005 Acrodermatitis continua of Hallopeau (disorder) 784328000 Pustular psoriasis of palm of hand (disorder) 27520001 Pustular psoriasis of palms and soles (disorder) 239098009 Acropustulosis of infancy (disorder) 784327005 Pustular psoriasis of sole of foot (disorder) Rupioid psoriasis (disorder) | 238617008 | Circinate and annular pustular psoriasis (disorder) |
| 238613007 Generalized pustular psoriasis of pregnancy (disorder) 238616004 Infantile pustular psoriasis (disorder) 238615000 Juvenile pustular psoriasis (disorder) 28840001 Generalized pustular psoriasis, exanthematous type (disorder) 238611009 Lapiere type of psoriasis (disorder) 81271001 Localized pustular psoriasis (disorder) 83839005 Acrodermatitis continua of Hallopeau (disorder) 784328000 Pustular psoriasis of palm of hand (disorder) 27520001 Pustular psoriasis of palms and soles (disorder) 239098009 Acropustulosis of infancy (disorder) 784327005 Pustular psoriasis of sole of foot (disorder) 200969003 Rupioid psoriasis (disorder) | 238612002 | Generalized pustular psoriasis (disorder) |
| 238616004Infantile pustular psoriasis (disorder)238615000Juvenile pustular psoriasis (disorder)28840001Generalized pustular psoriasis, exanthematous type (disorder)238611009Lapiere type of psoriasis (disorder)81271001Localized pustular psoriasis (disorder)83839005Acrodermatitis continua of Hallopeau (disorder)784328000Pustular psoriasis of palm of hand (disorder)27520001Pustular psoriasis of palms and soles (disorder)239098009Acropustulosis of infancy (disorder)784327005Pustular psoriasis of sole of foot (disorder)200969003Rupioid psoriasis (disorder) | 402326008 | Acute generalized pustular psoriasis de novo (disorder) |
| Juvenile pustular psoriasis (disorder) 28840001 Generalized pustular psoriasis, exanthematous type (disorder) 238611009 Lapiere type of psoriasis (disorder) 81271001 Localized pustular psoriasis (disorder) 83839005 Acrodermatitis continua of Hallopeau (disorder) 784328000 Pustular psoriasis of palm of hand (disorder) 27520001 Pustular psoriasis of palms and soles (disorder) 239098009 Acropustulosis of infancy (disorder) 784327005 Pustular psoriasis of sole of foot (disorder) 200969003 Rupioid psoriasis (disorder) | 238613007 | Generalized pustular psoriasis of pregnancy (disorder) |
| 28840001 Generalized pustular psoriasis, exanthematous type (disorder) 238611009 Lapiere type of psoriasis (disorder) 81271001 Localized pustular psoriasis (disorder) 83839005 Acrodermatitis continua of Hallopeau (disorder) 784328000 Pustular psoriasis of palm of hand (disorder) 27520001 Pustular psoriasis of palms and soles (disorder) 239098009 Acropustulosis of infancy (disorder) 784327005 Pustular psoriasis of sole of foot (disorder) 200969003 Rupioid psoriasis (disorder) | 238616004 | Infantile pustular psoriasis (disorder) |
| 238611009Lapiere type of psoriasis (disorder)81271001Localized pustular psoriasis (disorder)83839005Acrodermatitis continua of Hallopeau (disorder)784328000Pustular psoriasis of palm of hand (disorder)27520001Pustular psoriasis of palms and soles (disorder)239098009Acropustulosis of infancy (disorder)784327005Pustular psoriasis of sole of foot (disorder)200969003Rupioid psoriasis (disorder) | 238615000 | Juvenile pustular psoriasis (disorder) |
| 81271001Localized pustular psoriasis (disorder)83839005Acrodermatitis continua of Hallopeau (disorder)784328000Pustular psoriasis of palm of hand (disorder)27520001Pustular psoriasis of palms and soles (disorder)239098009Acropustulosis of infancy (disorder)784327005Pustular psoriasis of sole of foot (disorder)200969003Rupioid psoriasis (disorder) | 28840001 | Generalized pustular psoriasis, exanthematous type (disorder) |
| Acrodermatitis continua of Hallopeau (disorder) Pustular psoriasis of palm of hand (disorder) Pustular psoriasis of palms and soles (disorder) Pustular psoriasis of palms and soles (disorder) Acropustulosis of infancy (disorder) Pustular psoriasis of sole of foot (disorder) Pustular psoriasis (disorder) Rupioid psoriasis (disorder) | 238611009 | Lapiere type of psoriasis (disorder) |
| 784328000 Pustular psoriasis of palm of hand (disorder) 27520001 Pustular psoriasis of palms and soles (disorder) 239098009 Acropustulosis of infancy (disorder) 784327005 Pustular psoriasis of sole of foot (disorder) 200969003 Rupioid psoriasis (disorder) | 81271001 | Localized pustular psoriasis (disorder) |
| 27520001 Pustular psoriasis of palms and soles (disorder) 239098009 Acropustulosis of infancy (disorder) 784327005 Pustular psoriasis of sole of foot (disorder) 200969003 Rupioid psoriasis (disorder) | 83839005 | Acrodermatitis continua of Hallopeau (disorder) |
| 239098009 Acropustulosis of infancy (disorder) 784327005 Pustular psoriasis of sole of foot (disorder) 200969003 Rupioid psoriasis (disorder) | 784328000 | Pustular psoriasis of palm of hand (disorder) |
| 784327005 Pustular psoriasis of sole of foot (disorder) 200969003 Rupioid psoriasis (disorder) | 27520001 | Pustular psoriasis of palms and soles (disorder) |
| 200969003 Rupioid psoriasis (disorder) | 239098009 | Acropustulosis of infancy (disorder) |
| | 784327005 | Pustular psoriasis of sole of foot (disorder) |
| 238608008 Scalp psoriasis (disorder) | 200969003 | Rupioid psoriasis (disorder) |
| | 238608008 | Scalp psoriasis (disorder) |

| 25847004 | Seborrheic psoriasis (disorder) |
|---|---|
| 238601002 | Unstable psoriasis (disorder) |
| 161562002 | History of psoriasis (situation) |
| 11188005 | Psoriasiform napkin eruption (disorder) |
| 400069004 | Nevoid psoriasis (disorder) |
| 866341000000101 | Psoriasis area and severity index score (observable entity) |
| 239803008 | Juvenile psoriatic arthritis with psoriasis (disorder) |
| Contact Dermatitis | Juvernie psoriatic artifitis with psoriasis (disorder) |
| Read V2 Code | Code description |
| Myu21 | [X]Allergic contact dermatitis due to other chemical products |
| Myu23 | [X]Allergic contact dermatitis due to other agents |
| Myu24 | [X]Irritant contact dermatitis due to other chemical products |
| Myu25 | [X]Irritant contact dermatitis due to other agents |
| Myu26 | [X]Unspecified contact dermatitis due to other chemical products |
| Myu27 | [X]Unspecified contact dermatitis due to other agents |
| M12 | Contact dermatitis and other eczemas |
| M120. | Contact dermatitis due to detergents |
| M121. | Contact dermatitis due to oils and greases |
| M122. | Contact dermatitis due to solvents |
| M1220 | Contact dermatitis due to chlorocompound |
| M1221 | Contact dermatitis due to cyclohexane |
| M1222 | Contact dermatitis due to ester |
| M1223 | Contact dermatitis due to glycol |
| M1224 | Contact dermatitis due to hydrocarbon |
| M1225 | Contact dermatitis due to ketone |
| M122z | Contact dermatitis due to solvent NOS |
| M123. | Contact dermatitis due to drugs and medicaments |
| M1230 | Contact dermatitis due to arnica |
| M1231 | Contact dermatitis due to fungicides |
| M1232 | Contact dermatitis due to iodine |
| M1233 | Contact dermatitis due to keratolytics |
| M1234 | Contact dermatitis due to mercurials |
| M1235 | Contact dermatitis due to neomycin |
| M1236 | Contact dermatitis due to pediculocides |
| M1237 | Contact dermatitis due to phenols |
| M1238 | Contact dermatitis due to scabicides |
| M123z | Contact dermatitis due to medicament NOS |
| M124. | Contact dermatitis due to other chemical products |
| M1240 | Contact dermatitis due to acids |
| M1241 | Contact dermatitis due to adhesive plaster |
| M1242 | Contact dermatitis due to alkalis |
| M1243 | Contact dermatitis due to caustics |
| M1244 | Contact dermatitis due to dichromate |
| M1245 | Contact dermatitis due to insecticide |
| M1246 | Contact dermatitis due to nylon |
| M1247 | Contact dermatitis due to plastic |
| M1248 | Contact dermatitis due to rubber |

| M124z | Contact dermatitis: other chemicals NOS |
|---|---|
| M125. | Contact dermatitis due to food in contact with skin |
| M1250 | Contact dermatitis due to cereals |
| M1251 | Contact dermatitis due to fish |
| M1252 | Contact dermatitis due to flour |
| M1253 | Contact dermatitis due to fruit |
| M1254 | Contact dermatitis due to meat |
| M1255 | Contact dermatitis due to milk |
| M125z | Contact dermatitis due to food NOS |
| M126. | Contact dermatitis due to plants |
| M1260 | Contact dermatitis due to lacquer tree |
| M1261 | Contact dermatitis due to poison-ivy |
| M1262 | Contact dermatitis due to poison-oak |
| M1263 | Contact dermatitis due to poison-sumac |
| M1264 | Contact dermatitis due to poison-vine |
| M1265 | Contact dermatitis due to primrose |
| M1266 | Contact dermatitis due to ragweed |
| M126z | Contact dermatitis due to plants NOS |
| M128. | Allergic contact dermatitis |
| M1280 | Allergic contact dermatitis due to adhesives |
| M1281 | Allergic contact dermatitis due to cosmetics |
| M1282 | Allergic contact dermatitis due to drugs in contact with the skin |
| M1283 | Allergic contact dermatitis due to dyes |
| M1284 | Allergic contact dermatitis due to other chemical products |
| M1285 | Allergic contact dermatitis due to food in contact with the skin |
| M1286 | Allergic contact dermatitis due to plants, except food |
| M129. | Irritant contact dermatitis |
| M1290 | Irritant contact dermatitis due to cosmetics |
| M1291 | Irritant contact dermatitis due to drugs in contact with the skin |
| M1292 | Irritant contact dermatitis due to other chemical products |
| M1293 | Irritant contact dermatitis due to food in contact with the skin |
| M1294 | Irritant contact dermatitis due to plants, except food |
| M12y. | Contact dermatitis due to other specified agents |
| M12y0 | Contact dermatitis due to other specified agents Contact dermatitis due to cosmetics |
| • | Contact dermatitis due to cosmetics Contact dermatitis due to cold weather |
| M12y1 | Contact dermatitis due to dyes |
| M12y2 | Contact dermatitis due to dyes Contact dermatitis due to furs |
| M12y3 | |
| M12y4 | Contact dermatitis due to hot weather |
| M12y5 | Contact dermatitis due to infra-red rays |
| M12y6 | Contact dermatitis due to jewellery |
| M12y7 | Contact dermatitis due to light (excluding sunlight) |
| M12y8 | Contact dermatitis due to metals |
| M12y9 | Contact dermatitis due to preservatives |
| M12yA | Contact dermatitis due to radiation NOS |
| M12yB | Contact dermatitis due to ultra-violet rays (excluding sunlight) |
| M12yC | Contact dermatitis due to x-rays |
| M12yD | Contact dermatitis due to casting materials |

| M12yz | Contact dermatitis: specified agent NOS |
|---|---|
| M12z. | Contact dermatitis NOS |
| M12zz | Contact dermatitis NOS |
| Read CTV3 Code | Description |
| Xa9CV | Contact dermatitis |
| X505x | Allergic contact dermatitis |
| X505y | Nickel sensitivity |
| X505z | Implant allergic nickel contact dermatitis |
| X5060 | Ingested allergen contact dermatitis |
| Xa0Wg | Baboon syndrome |
| X5061 | Photoallergic contact dermatitis |
| M1280 | |
| | Allergic contact dermatitis due to adhesives |
| M1281 | Allergic contact dermatitis due to cosmetics |
| M1282 | Allergic contact dermatitis due to drugs in contact with the skin |
| M1283 | Allergic contact dermatitis due to dyes |
| M1284 | Allergic contact dermatitis due to other chemical products |
| M1285 | Allergic contact dermatitis due to food in contact with the skin |
| M1286 | Allergic contact dermatitis due to plants, except food |
| Myu21 | [X]Allergic contact dermatitis due to other chemical products |
| Myu23 | [X]Allergic contact dermatitis due to other agents |
| X5063 | Irritant contact dermatitis |
| X5040 | Fibreglass dermatitis |
| X5064 | Acute irritant contact dermatitis |
| X5065 | Subacute irritant contact dermatitis |
| X5066 | Chronic irritant contact dermatitis |
| Xa0WJ | Swimming pool dermatitis |
| X505H | Cactus dermatitis |
| Xa13g | Coral dermatitis |
| M123. | Drug-induced contact dermatitis |
| M1230 | Contact dermatitis due to arnica |
| M1231 | Contact dermatitis due to fungicides |
| M1232 | Contact dermatitis due to iodine |
| M1233 | Contact dermatitis due to keratolytics |
| M1234 | Contact dermatitis due to mercurials |
| M1235 | Contact dermatitis due to neomycin |
| M1236 | Contact dermatitis due to pediculocides |
| M1237 | Contact dermatitis due to phenols |
| M1238 | Contact dermatitis due to scabicides |
| M123z | Contact dermatitis due to medicament NOS |
| M1290 | Irritant contact dermatitis due to cosmetics |
| M1291 | Irritant contact dermatitis due to drugs in contact with the skin |
| M1292 | Irritant contact dermatitis due to other chemical products |
| M1293 | Irritant contact dermatitis due to food in contact with the skin |
| M1294 | Irritant contact dermatitis due to plants, except food |
| Myu24 | [X]Irritant contact dermatitis due to other chemical products |
| Myu25 | [X]Irritant contact dermatitis due to other agents |
| X5062 | Occupational allergic contact dermatitis |

| XE1Ar | Contact dermatitis due to adhesive plaster |
|-------|------------------------------------------------------|
| X505t | Elastoplast contact dermatitis |
| M120. | Contact dermatitis due to detergents |
| M122. | Contact dermatitis due to solvents |
| M1220 | Contact dermatitis due to chlorocompound |
| M1221 | Contact dermatitis due to cyclohexane |
| M1222 | Contact dermatitis due to ester |
| M1223 | Contact dermatitis due to glycol |
| M1224 | Contact dermatitis due to hydrocarbon |
| M1225 | Contact dermatitis due to ketone |
| M122z | Contact dermatitis due to solvent NOS |
| M124. | Contact dermatitis due to other chemical products |
| M1240 | Contact dermatitis due to acids |
| M1242 | Contact dermatitis due to alkalis |
| M1243 | Contact dermatitis due to caustics |
| M1244 | Contact dermatitis due to dichromate |
| M1245 | Contact dermatitis due to insecticide |
| M1246 | Contact dermatitis due to nylon |
| M1247 | Contact dermatitis due to plastic |
| M1248 | Contact dermatitis due to rubber |
| M124z | Contact dermatitis: other chemicals NOS |
| M125. | Contact dermatitis due to food in contact with skin |
| M1250 | Contact dermatitis due to cereals |
| M1251 | Contact dermatitis due to fish |
| M1252 | Contact dermatitis due to flour |
| M1253 | Contact dermatitis due to fruit |
| M1254 | Contact dermatitis due to meat |
| M1255 | Contact dermatitis due to milk |
| X505u | Egg contact dermatitis |
| XE1As | Contact dermatitis due to food NOS |
| M126. | Contact dermatitis due to plants |
| M1260 | Contact dermatitis due to lacquer tree |
| M1261 | Contact dermatitis due to poison-ivy |
| M1262 | Contact dermatitis due to poison-oak |
| M1263 | Contact dermatitis due to poison-sumac |
| M1264 | Contact dermatitis due to poison-vine |
| M1265 | Contact dermatitis due to primrose |
| M1266 | Contact dermatitis due to ragweed |
| M126z | Contact dermatitis due to plants NOS |
| M12y. | Contact dermatitis due to other specified agents |
| M12y1 | Contact dermatitis due to cold weather |
| M12y2 | Contact dermatitis due to dyes |
| M12y3 | Contact dermatitis due to furs |
| M12y4 | Contact dermatitis due to hot weather |
| M12y5 | Contact dermatitis due to infrared rays |
| M12y6 | Contact dermatitis due to jewellery |
| M12y7 | Contact dermatitis due to light (excluding sunlight) |

| Contact dermatitis due to preservatives |
|------------------------------------------------------------------|
| Contact dermatitis due to radiation NOS |
| Contact dermatitis due to ultraviolet rays (excluding sunlight) |
| Contact dermatitis due to X-rays |
| Contact dermatitis due to casting materials |
| Contact dermatitis: specified agent NOS |
| Lanolin contact dermatitis |
| Contact dermatitis due to cosmetics |
| Perfume contact dermatitis |
| Contact dermatitis due to metals |
| Contact dermatitis NOS |
| [X]Unspecified contact dermatitis due to other chemical products |
| [X]Unspecified contact dermatitis due to other agents |
| Contact dermatitis due to oils and greases |
| Grease contact dermatitis |
| Oil contact dermatitis |
| Contact dermatitis - chemicals |
| Contact dermatitis - foods/plants |
| Description |
| Irritant contact dermatitis caused by detergent (disorder) |
| Irritant contact dermatitis caused by rubber |
| Irritant contact dermatitis caused by chemical (disorder) |
| Irritant contact dermatitis caused by metal (disorder) |
| Allergic contact dermatitis caused by latex (disorder) |
| Allergic contact dermatitis caused by plant material (disorder) |
| Allergic contact dermatitis caused by pollen (disorder) |
| Allergic contact dermatitis caused by chemical (disorder) |
| Contact dermatitis of right upper and lower eyelids (disorder) |
| Contact dermatitis caused by poison sumac (disorder) |
| Irritant contact dermatitis (disorder) |
| Acute contact dermatitis (disorder) |
| Contact dermatitis caused by phenol (disorder) |
| Contact dermatitis due to other drug, NEC (disorder) |
| Contact dermatitis caused by insecticide |
| Contact dermatitis due to other non food plant (disorder) |
| Contact dermatitis due to other specified agents (disorder) |
| Photoallergic contact dermatitis |
| Contact dermatitis caused by solar radiation (disorder) |
| Contact dermatitis of bilateral lower eyelids |
| Generalized exfoliative contact dermatitis (disorder) |
| Contact dermatitis caused by adhesive bandage (disorder) |
| Contact dermatitis due to fur (disorder) |
| Urine-induced contact dermatitis (disorder) |
| Contact dermatitis/eczema |
| Contact dermatitis due to detergents (disorder) |
| Contact dermatitis due to oils and greases (disorder) |

| 156342007 | Drug-induced contact dermatitis (disorder) |
|---|---|
| 156343002 | Contact dermatitis: [chemicals] or [elastoplast allergy] |
| 156344008 | Contact dermatitis - foods/plants (disorder) |
| 156345009 | (Contact dermatitis: sun) or (Farmers skin) or (photosensitivity - sun) or (sunburn) (disorder) |
| 156346005 | Contact dermatitis: metals(& [nickel]) (disorder) |
| 156348006 | (Contact dermatitis NOS) or (discoid eczema) or (nummular eczema) (disorder) |
| 15681161000119107 | Contact dermatitis of bilateral eyelids (disorder) |
| 16228891000119105 | Allergic contact dermatitis caused by metal (disorder) |
| 17946007 | Contact dermatitis caused by fungicide (disorder) |
| 18793008 | Contact dermatitis caused by fruit (disorder) |
| 193918001 | Contact &/or allergic eyelid dermatitis (disorder) (Contact dermatitis [& other eczemas]) or (contact eczema) or (occupational dermatitis) (disorder) |
| 200781007 | Contact dermatitis due to detergents (disorder) |
| 200782000 | Contact dermatitis due to oils &/or greases (disorder) |
| 200783005 | Contact dermatitis due to solvents (disorder) |
| 200784004 | Contact dermatitis caused by chlorocompound |
| 200785003 | Contact dermatitis caused by cyclohexane group |
| 200786002 | Contact dermatitis caused by ester (disorder) |
| 200787006 | Contact dermatitis caused by glycol |
| 200788001 | Contact dermatitis caused by hydrocarbon (disorder) |
| 200789009 | Contact dermatitis caused by ketone (disorder) |
| 200790000 | Contact dermatitis due to solvent NOS (disorder) |
| 200791001 | Contact dermatitis due to arnica (disorder) |
| 200792008 | Contact dermatitis due to fungicides (disorder) |
| 200793003 | Contact dermatitis due to iodine (disorder) |
| 200794009 | Contact dermatitis caused by keratolytic |
| 200795005 | Contact dermatitis due to mercurials (disorder) |
| 200796006 | Contact dermatitis due to neomycin (disorder) |
| 200797002 | Contact dermatitis due to pediculicides (disorder) |
| 200798007 | Contact dermatitis due to phenols (disorder) |
| 200799004 | Contact dermatitis due to scabicides (disorder) |
| 200800000 | Contact dermatitis due to medicament NOS (disorder) |
| 200801001 | Contact dermatitis due to other chemical products (disorder) |
| 200802008 | Contact dermatitis caused by acid (disorder) |
| 200803003 | Contact dermatitis due to adhesive plaster (& elastoplast) (disorder) |
| 200804009 | Contact dermatitis caused by alkali (disorder) |
| 200805005 | Contact dermatitis due to caustic |
| 200806006 | Contact dermatitis due to dichromate (disorder) |
| 200807002 | Contact dermatitis due to insecticide (disorder) |
| 200808007 | Contact dermatitis due to nylon (disorder) |
| 200809004 | Contact dermatitis due to plastic (disorder) |
| 200810009 | Contact dermatitis due to rubber (disorder) |
| 200811008 | Contact dermatitis: other chemicals NOS (disorder) |
| 200813006 | Contact dermatitis due to food in contact with skin (disorder) |
| 200814000 | Contact dermatitis due to cereals (disorder) |

| | <del>,</del> |
|---|---|
| 200815004 | Contact dermatitis due to fish (disorder) |
| 200816003 | Contact dermatitis due to flour (disorder) |
| 200817007 | Contact dermatitis due to fruit (disorder) |
| 200818002 | Contact dermatitis due to meat (disorder) |
| 200819005 | Contact dermatitis due to milk (disorder) |
| 200820004 | (Contact dermatitis due to food NOS) or (egg contact dermatitis) (disorder) |
| 200821000 | Contact dermatitis caused by plants |
| 200822007 | Contact dermatitis due to lacquer tree (disorder) |
| 200823002 | Contact dermatitis caused by poison ivy (disorder) |
| 200824008 | Contact dermatitis caused by poison oak |
| 200825009 | Contact dermatitis due to poison-sumac (disorder) |
| 200826005 | Contact dermatitis due to poison-vine (disorder) |
| 200827001 | Contact dermatitis due to primrose (disorder) |
| 200828006 | Contact dermatitis due to ragweed (disorder) |
| 200829003 | Contact dermatitis due to plants NOS (disorder) |
| 200830008 | Contact dermatitis due to solar radiation (disorder) |
| 200831007 | Unspecified contact dermatitis due to solar radiation (disorder) |
| 200836002 | Photocontact dermatitis |
| 200840006 | Contact dermatitis due to solar radn NOS (disorder) |
| 200841005 | Allergic contact dermatitis (disorder) |
| 200842003 | Allergic contact dermatitis due to adhesive |
| 200843008 | Allergic contact dermatitis due to cosmetic |
| 200844002 | Allergic contact dermatitis due to drug in contact with skin |
| 200845001 | Allergic contact dermatitis due to dye |
| 200846000 | Allergic contact dermatitis due to other chemical products (disorder) |
| 200847009 | Allergic contact dermatitis caused by food in contact with skin |
| 200848004 | Allergic contact dermatitis caused by plants, except food (disorder) |
| 200850007 | Irritant contact dermatitis (disorder) |
| 200851006 | Irritant contact dermatitis due to cosmetic |
| 200852004 | Irritant contact dermatitis due to drug in contact with skin |
| 200853009 | Irritant contact dermatitis due to other chemical products (disorder) |
| 200854003 | Irritant contact dermatitis due to food in contact with skin |
| 200855002 | Irritant contact dermatitis caused by plants, except food (disorder) |
| 200867000 | Contact dermatitis due to other specified agents (disorder) |
| 200869002 | Contact dermatitis due to cold weather (disorder) |
| 200870001 | Contact dermatitis due to dyes (disorder) |
| 200871002 | Contact dermatitis due to fur |
| 200872009 | Contact dermatitis due to hot weather (disorder) |
| 200873004 | Contact dermatitis due to infrared rays (disorder) |
| 200874005 | Contact dermatitis due to immarca rays (disorder) |
| 200875006 | Contact dermatitis due to light (excluding sunlight) (disorder) |
| 200876007 | (Contact dermatitis due to metals) or (nickel sensitivity) (disorder) |
| 200877003 | Contact dermatitis due to inetals of (inetel sensitivity) (disorder) |
| 200878008 | Contact dermatitis due to radiation NOS (disorder) |
| 200879000 | Contact dermatitis due to radiation Nos (disorder) Contact dermatitis caused by ultraviolet rays (excluding sunlight) |
| 200879000 | Contact dermatitis due to X-rays (disorder) |
| 200881003 | Contact dermatitis due to X-rays (disorder) Contact dermatitis caused by casting materials |
| 200001003 | Contact defination caused by casting materials |

| 200882005 | Contact dermatitis: specified agent NOS (disorder) |
|---|---|
| 200883000 | Contact dermatitis NOS (disorder) |
| 200889001 | Contact dermatitis NOS (disorder) |
| 201360000 | [X]Allergic contact dermatitis due to other chemical products (disorder) |
| 201361001 | [X]Allergic contact dermatitis due to other agents (disorder) |
| 201362008 | [X]Irritant contact dermatitis due to other chemical products (disorder) |
| 201363003 | [X]Irritant contact dermatitis due to other agents (disorder) |
| 201364009 | [X]Unspecified contact dermatitis due to other chemical products (disorder) |
| 201365005 | [X]Unspecified contact dermatitis due to other agents (disorder) |
| 22131007 | Contact dermatitis due to ultraviolet rays, except sun (disorder) |
| 22353002 | Contact dermatitis due to glycol group (disorder) |
| 23012005 | Contact dermatitis caused by solvents |
| 238506004 | Contact dermatitis due to cold weather |
| 238524002 | Photoallergic contact dermatitis |
| 238568000 | Grease contact dermatitis (disorder) |
| 238569008 | Oil contact dermatitis (disorder) |
| 238570009 | Elastoplast contact dermatitis (disorder) |
| 238571008 | Egg contact dermatitis (disorder) |
| 238572001 | Lanolin contact dermatitis (disorder) |
| 238573006 | Perfume contact dermatitis (disorder) |
| 238575004 | Allergic contact dermatitis (disorder) |
| 238576003 | Allergic contact dermatitis caused by nickel implant (disorder) |
| 238577007 | Ingested allergen contact dermatitis (disorder) |
| 238578002 | Occupational allergic contact dermatitis (disorder) |
| 238579005 | Acute irritant contact dermatitis (disorder) |
| 238580008 | Subacute irritant contact dermatitis (disorder) |
| 238581007 | Chronic irritant contact dermatitis (disorder) |
| 238583005 | Saliva-induced contact dermatitis (disorder) |
| 238584004 | Feces-induced contact dermatitis (disorder) |
| 238672005 | Lichenoid allergic contact dermatitis (disorder) |
| 247469006 | Urine-induced contact dermatitis (disorder) |
| 25664003 | Contact dermatitis due to dichlorvos |
| 26208004 | Contact dermatitis due to keratolytic agent (disorder) |
| 26532007 | Contact dermatitis caused by scabicide (disorder) |
| 267648006 | Contact or allergic eyelid dermatitis (disorder) |
| 267792000 | Contact dermatitis and other eczemas (disorder) |
| 267793005 | Contact dermatitis due to oil and grease |
| 267794004 | Contact dermatitis due to food NOS (disorder) |
| 267795003 | Contact dermatitis due to cosmetics (disorder) |
| 267796002 | Contact dermatitis due to metal (disorder) |
| | Contact dermatitis/eczema (& [allergic eczema - extrinsic] or [occupational |
| 267842005 | eczema]) |
| 267843000 | Contact dermatitis: [chemicals] or [elastoplast allergy] |
| 267844006 | (Contact dermatitis: sun) or (Farmers skin) or (photosensitivity - sun) or (sunburn) (disorder) |
| 267845007 | Contact dermatitis: metals(& [nickel]) (disorder) |
| 279334008 | Contact dermatitis due to infra-red rays |
| 287003002 | Contact dermatitis - chemicals (disorder) |

| 287004008 | Contact dermatitis - foods/plants (disorder) |
|---|---|
| 2889003 | Contact dermatitis due to alkali (disorder) |
| 291000119100 | Contact dermatitis caused by chemical (disorder) |
| 30451004 | Contact dermatitis due to detergent |
| 31948006 | Contact dermatitis caused by plastic (disorder) |
| 3226008 | Contact dermatitis - chemicals |
| 32371003 | Contact dermatitis caused by neomycin (disorder) |
| 342761000119104 | Allergic contact dermatitis of right upper eyelid (disorder) |
| 342771000119105 | Allergic contact dermatitis of right lower eyelid |
| 342781000119108 | Allergic contact dermatitis of right eyelid (disorder) |
| 342791000119106 | Allergic contact dermatitis of left upper eyelid |
| 342801000119107 | Allergic contact dermatitis of left lower eyelid (disorder) |
| 342811000119105 | Allergic contact dermatitis of left eyelid (disorder) |
| 36530008 | Contact dermatitis caused by fish |
| 39670009 | Contact dermatitis due to chlorocompound group (disorder) |
| 402249007 | Allergic contact dermatitis of eyelid |
| 402252004 | Allergic contact dermatitis of perianal skin |
| 402253009 | Allergic contact dermatitis of external ear |
| 402254003 | Allergic contact dermatitis of hands |
| 402255002 | Allergic contact dermatitis of lower leg |
| 402256001 | Allergic contact dermatitis of male genitalia |
| 402257005 | Allergic contact dermatitis of female genitalia |
| 402261004 | Acute irritant contact dermatitis |
| 402263001 | Cumulative irritant contact dermatitis of hands caused by wet work |
| 402265008 | Irritant contact dermatitis of hands caused by oil and/or grease (disorder) |
| 402266009 | Irritant contact dermatitis of hands caused by solvent |
| 402267000 | Irritant contact dermatitis caused by metal swarf (disorder) |
| 402268005 | Irritant contact dermatitis caused by cement (disorder) |
| 402269002 | Irritant contact dermatitis of hands caused by cement (disorder) |
| 402270001 | Irritant contact dermatitis of hands caused by friction |
| 402271002 | Irritant contact dermatitis caused by chlorine |
| 402272009 | Irritant contact dermatitis caused by biocide (disorder) |
| 402273004 | Cumulative irritant contact dermatitis of hands |
| 402274005 | Cumulative irritant contact dermatitis |
| | Irritant contact dermatitis caused by contact with urine and/or feces |
| 402275006 | (disorder) |
| 402276007 | Irritant contact dermatitis due to incontinence |
| 402278008 | Irritant contact dermatitis due to stoma/fistula |
| 402279000 | Irritant contact dermatitis due to ileostomy |
| 402280002 | Irritant contact dermatitis due to colostomy |
| 402281003 | Irritant contact dermatitis due to urostomy |
| 402284006 | Irritant contact dermatitis due to dribbling and/or teething |
| 402290005 | Irritant contact hand dermatitis |
| 402291009 | Contact dermatitis of hands |
| 402577002 | Allergic contact dermatitis by site |
| 402578007 | Irritant contact dermatitis caused by detergent and/or wet work (disorder) |
| 402579004 | Irritant contact dermatitis caused by plant |

| 402580001 | Irritant contact dermatitis caused by oil and/or grease (disorder) |
|---|---|
| 402581002 | Irritant contact dermatitis caused by wood (disorder) |
| 402582009 | Irritant contact dermatitis caused by solvent (disorder) |
| 402584005 | Occupational irritant contact dermatitis |
| 40275004 | Contact dermatitis and other eczemas |
| 403585004 | Contact psychodermatitis |
| 405244005 | Urine induced contact dermatitis |
| 40712008 | Contact dermatitis caused by arnica |
| 409784006 | Contact dermatitis caused by Rhus diversiloba (disorder) |
| 409785007 | Contact dermatitis caused by Rhus quercifolia |
| 410049000 | Contact dermatitis caused by Genus Toxicodendron |
| 419121001 | Allergic contact dermatitis of pinna |
| 419957005 | Allergic contact dermatitis of external auditory canal |
| 42409002 | Contact dermatitis due to oils (disorder) |
| 425630003 | Acute irritant contact dermatitis |
| 42733007 | Contact dermatitis caused by dichromate |
| 44210006 | Contact dermatitis due to preservative (disorder) |
| 45309006 | Allergic contact dermatitis caused by secretions (disorder) |
| 46240005 | Contact dermatitis caused by rubber (disorder) |
| 46787004 | Contact dermatitis caused by light, except sun (disorder) |
| 48681004 | Contact dermatitis due to hot weather (disorder) |
| 49186001 | Contact dermatitis caused by cereal (disorder) |
| 51221005 | Chronic contact dermatitis (disorder) |
| 51732009 | Contact dermatitis due to hydrocarbon group (disorder) |
| 5205006 | Contact dermatitis due to poison ivy (disorder) |
| 5221001 | Contact dermatitis due to greases (disorder) |
| 52811009 | Contact dermatitis due to ketone group (disorder) |
| 53930004 | Contact dermatitis caused by ragweed (disorder) |
| 55113003 | Contact dermatitis due to poison oak (disorder) |
| 55934006 | Contact dermatitis caused by flour |
| 56669003 | Contact dermatitis due to ester group (disorder) |
| 586008 | Contact dermatitis caused by primrose (disorder) |
| 58843002 | Contact dermatitis due to caustic agent (disorder) |
| 59336008 | Contact dermatitis due to cold weather (disorder) |
| 64451001 | Contact dermatitis due to cyclohexane group (disorder) |
| 65129009 | Contact dermatitis caused by milk |
| 65394002 | Contact dermatitis caused by Rhus verniciflua |
| 67445002 | Contact dermatitis caused by food in contact with skin (disorder) |
| 67607005 | Contact dermatitis due to infrared rays (disorder) |
| 68670009 | Contact dermatitis of eyelid (disorder) |
| 6888008 | Contact dermatitis caused by dye (disorder) |
| 69827001 | Contact dermatitis due to X-ray |
| 69999007 | Contact dermatitis caused by plants, except food |
| 700340008 | Allergic contact dermatitis of upper eyelid (disorder) |
| 700341007 | Allergic contact dermatitis of lower eyelid |
| 715150009 | Contact dermatitis caused by Senecio jacobea |

| 717725000 | Contact dermatitis of female genitalia |
|---|---|
| 72057009 | Contact dermatitis caused by pediculicide |
| 724635009 | Contact dermatitis of external ear |
| 724825001 | Allergic contact dermatitis caused by hairdressing product (disorder) |
| 724828004 | Irritant contact dermatitis caused by cosmetic substance |
| 724829007 | Occupational contact dermatitis |
| 724869008 | Protein contact dermatitis |
| 72921001 | Contact dermatitis caused by meat |
| 733201000 | Irritant contact dermatitis caused by dietary substance (disorder) |
| 735758003 | Irritant contact dermatitis caused by friction |
| 735759006 | Irritant contact dermatitis caused by sweat |
| 735760001 | Irritant contact dermatitis caused by body fluid |
| 762379000 | Allergic contact dermatitis caused by dental material (disorder) |
| 762380002 | Allergic contact dermatitis caused by food flavour |
| 762381003 | Allergic contact dermatitis caused by food additive (disorder) |
| 762382005 | Allergic contact dermatitis caused by agrochemical biocide |
| 762383000 | Allergic contact dermatitis caused by agrocinemical blockde |
| | Allergic contact dermatitis caused by disinfectant (disorder) |
| 762384006 | Allergic contact dermatitis caused by distrilectant (disorder) Allergic contact dermatitis caused by allergenic hapten derived from plants |
| 762385007 | or organic matter |
| 762386008 | Allergic contact dermatitis caused by rubber compound |
| 762387004 | Allergic contact dermatitis caused by systemic medicament |
| 762388009 | Irritant contact dermatitis caused by emollient substance (disorder) |
| 762545002 | Occupational allergic contact dermatitis caused by footwear (disorder) |
| 762548000 | Occupational allergic contact dermatitis caused by cosmetic |
| 762549008 | Occupational allergic contact dermatitis caused by fragrance |
| 762552000 | Occupational allergic contact dermatitis caused by dental material |
| 762554004 | Occupational allergic contact dermatitis caused by food flavor |
| 762555003 | Occupational allergic contact dermatitis caused by food additive (disorder) |
| | Occupational allergic contact dermatitis caused by hairdressing product |
| 762558001 | (disorder) |
| 762560004 | Occupational allergic contact dermatitis caused by agrochemical biocide (disorder) |
| 762561000 | Occupational allergic contact dermatitis caused by cutting oil |
| 762562007 | Occupational allergic contact dermatitis caused by disinfectant (disorder) |
| 762566005 | Occupational allergic contact dermatitis caused by metal compound |
| | Occupational allergic contact dermatitis caused by allergenic hapten derived |
| 762568006 | from plant (disorder) Occupational allergic contact dermatitis caused by industrial preservative |
| 762570002 | (disorder) |
| 762571003 | Occupational allergic contact dermatitis caused by biocide |
| 762574006 | Occupational allergic contact dermatitis caused by rubber compound |
| 702374000 | Occupational allergic contact dermatitis caused by systemic drug or |
| 762576008 | medicament |
| | Occupational allergic contact dermatitis caused by topical medicament |
| 762578009 | (disorder) |
| 762726008 | Occupational allergic contact dermatitis caused by clothing |
| 762754001 | Allergic contact dermatitis caused by fragrance (disorder) |
| 762755000 | Allergic contact dermatitis caused by footwear (disorder) |
| 762757008 | Allergic contact dermatitis caused by clothing |

| 76982008 | Contact dermatitis due to neicen vine |
|---|---|
| 770545005 | Contact dermatitis due to poison vine |
| 770588002 | Allergic contact dermatitis caused by iodine (disorder) Allergic contact dermatitis caused by iodophore (disorder) |
| 770588002 | Allergic contact dermatitis caused by louophore (disorder) Allergic contact dermatitis caused by povidone iodine (disorder) |
| 77560002 | Contact dermatitis due to adhesive plaster |
| 78079005 | <u> </u> |
| | Allergic contact dermatitis due to excretions Contact dermatitis due to metal |
| 78634007<br>78755001 | Contact dermatitis due to metal Contact dermatitis due to cosmetics |
| 788971005 | Irritant contact dermatitis of external ear (disorder) |
| 79927003 | Contact dermatitis due to acid (disorder) |
| 81351008 | Contact dermatitis due to acid (disorder) Contact dermatitis caused by radiation (disorder) |
| 81531008 | Contact dermatitis due to mercurials |
| | Contact dermatitis due to infercuriais Contact dermatitis due to iodine |
| 83150005<br>83508001 | Contact dermatitis due to hourse Contact dermatitis due to hylon |
| 85512009 | Contact dermatitis due to hylon Contact dermatitis due to jewellery |
| 86062001 | Contact dermatitis due to Jeweilery Contact dermatitis caused by drugs AND/OR medicine |
| 860924005 | Allergic contact dermatitis caused by alkali-metal soap (disorder) |
| 870749003 | Allergic contact dermatitis caused by assic acid (disorder) |
| 88718007 | Subacute contact dermatitis Subacute contact dermatitis |
| 91487003 | Urine-induced contact dermatitis |
| 93418006 | Contact dermatitis due to chromium |
| 93419003 | Contact dermatitis due to metals |
| 10762031000119106 | Contact dermatitis due to metals Contact dermatitis of left upper and lower eyelids (disorder) |
| Photodermatitis Photodermatitis | contact definitions of left apper and lower cyclias (disorder) |
| Read V2 Code | Code description |
| M1273 | Photodermatitis |
| M1274 | Photosensitiveness |
| | Photosensitiveness Photocontact dermatitis [berloque dermatitis] |
| M1274 | Photocontact dermatitis [berloque dermatitis] |
| M1274<br>M1278 | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme |
| M1274<br>M1278<br>M1279 | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response |
| M1274<br>M1278<br>M1279<br>M12A0 | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response |
| M1274 M1278 M1279 M12A0 M12A1 | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response |
| M1274 M1278 M1279 M12A0 M12A1 M1272 | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code M1273 | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description Photodermatitis |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code M1273 M1274 | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description Photodermatitis Photosensitivity of skin |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code M1273 M1274 X504r | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description Photodermatitis Photosensitivity of skin Photosensitisation reaction |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code M1273 M1274 X504r X504z | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description Photodermatitis Photosensitivity of skin Photosensitisation reaction Hydroa vacciniforme |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code M1273 M1274 X504r X504z X50Gr | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description Photodermatitis Photosensitivity of skin Photosensitisation reaction Hydroa vacciniforme Drug-induced photosensitivity |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code M1273 M1274 X504r X504z X50Gs | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description Photodermatitis Photosensitivity of skin Photosensitisation reaction Hydroa vacciniforme Drug-induced photosensitivity Drug phototoxic response |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code M1273 M1274 X504r X504r X50Gs X50Gs | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description Photodermatitis Photosensitivity of skin Photosensitivity of skin Hydroa vacciniforme Drug-induced photosensitivity Drug phototoxic response Drug photoallergic response |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code M1273 M1274 X504r X504r X50Gr X50Gs X50Gt Xa0Wh | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description Photodermatitis Photosensitivity of skin Photosensitisation reaction Hydroa vacciniforme Drug-induced photosensitivity Drug photoallergic response Drug-induced persistent light reaction |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code M1273 M1274 X504r X504r X50Gs X50Gs X50Gt Xa0Wh M1272 | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description Photodermatitis Photosensitivity of skin Photosensitisation reaction Hydroa vacciniforme Drug-induced photosensitivity Drug phototoxic response Drug photoallergic response Drug-induced persistent light reaction Hydroa aestivale |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code M1273 M1274 X504r X504r X50Gr X50Gs X50Gt Xa0Wh M1272 SNOMED CT ID | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description Photodermatitis Photosensitivity of skin Photosensitisation reaction Hydroa vacciniforme Drug-induced photosensitivity Drug phototoxic response Drug photoallergic response Drug-induced persistent light reaction Hydroa aestivale Description |
| M1274 M1278 M1279 M12A0 M12A1 M1272 Read CTV3 Code M1273 M1274 X504r X504r X504z X50Gr X50Gs X50Gt Xa0Wh M1272 SNOMED CT ID 111209006 | Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response Hydroa aestivale Description Photodermatitis Photosensitivity of skin Photosensitisation reaction Hydroa vacciniforme Drug-induced photosensitivity Drug photoallergic response Drug photoallergic response Drug-induced persistent light reaction Hydroa aestivale Description Photoallergic dermatitis |

| 200832000<br>200836002<br>200837006<br>200857005 | Hydroa aestivale Photocontact dermatitis [berloque dermatitis] Hydroa vacciniforme Drug phototoxic response Drug photoallergic response |
|---|---|
| 200837006<br>200857005 | Hydroa vacciniforme Drug phototoxic response |
| 200857005 | Drug phototoxic response |
| 200050000 | Drug photoallergic response |
| 200858000 | 01 0 1 |
| 201015007 | Hydroa aestivale |
| 22649008 | Photodermatitis |
| 238521005 | Plant photodermatitis |
| 238523008 | Photoallergic eczema |
| 238524002 | Photoallergic contact dermatitis |
| 238525001 | Polymorphic photodermatitis |
| 238527009 | Persistent light reaction |
| 259097007 | Delayed photoallergic dermatitis |
| 259608005 | Photodermatitis due to sun |
| 27687007 | Hydroa aestivale |
| 277805004 | Drug-induced persistent light reaction |
| 363619000 | Phototoxic phytotoxin |
| 367334003 | Photoallergic eczema |
| 367484009 | Photodermatitis due to sun |
| 402168004 | Acute phototoxic reaction (disorder) |
| 402172000 | Hypermelanosis due to phytophotodermatitis (disorder) |
| 402173005 | Phototoxic reaction to topical chemical (disorder) |
| 402174004 | Phototoxic reaction to dye (disorder) |
| 402175003 | Phototoxic reaction to tar or derivatives (disorder) |
| 402176002 | Phototoxic reaction to topically applied medicament (disorder) |
| 402480004 | Porphyria-induced phototoxic burn (disorder) |
| 44483004 | Phytophotodermatitis |
| 450907007 | Hydroa vacciniforme-like lymphoma (morphologic abnormality) |
| 45832002 | Pupil afferent light reaction |
| 53597009 | Phototoxic dermatitis |
| 58306008 | Acute phytophotodermatitis |
| 58419006 | Chronic phytophotodermatitis |
| 61064008 | Photodermatitis due to sun |
| 69231004 | Chronic phototoxic dermatitis |
| | Occupational phototoxic reaction to skin contact with exogenous |
| 724873006 | photoactive agent (disorder) |
| 737249005 | Photodermatitis co-occurrent and due to autoimmune disease (disorder) |
| 737250005 | Phototoxic reaction of skin caused by fragrance (disorder) |
| 737251009 | Phototoxic reaction of skin caused by cosmetic |
| 763719001 | Hydroa vacciniforme-like lymphoma (disorder) |
| 789440003 | Hydroa vacciniforme-like lymphoproliferative disorder |
| 80346008 | Drug photoallergic response |
| 83627000 | Drug phototoxic response |
| 84326006 | Phototoxicity |
| 95349002 | Phytophotodermatitis due to topical exposure to furocoumarin (disorder) |
| Ichthyosis | |
| Read V2 Code | Code description |

| M211. | Ichthyosis - acquired |
|----------------|-------------------------------------------------------|
| M2116 | Acquired ichthyosis |
| PH1 | Ichthyosis congenita |
| PH10. | Congenital ichthyosis, unspecified |
| PH11. | Harlequin fetus |
| PH12. | Ichthyosiform erythroderma |
| PH13. | Collodion baby |
| PH14. | Ichthyosis vulgaris |
| PH15. | X-linked ichthyosis |
| PH1y. | Other specified ichthyosis congenita |
| PH1y0 | Nethertons syndrome |
| PH1z. | Ichthyosis congenita NOS |
| Read CTV3 Code | Description |
| PH1 | Congenital ichthyosis |
| X78C8 | Ichthyosis vulgaris |
| X78C9 | Autosomal dominant ichthyosis vulgaris |
| X78CB | X-linked recessive ichthyosis |
| X78CA | Severe ichthyoses |
| PH13. | Lamellar ichthyosis |
| X78CD | Erythrodermic lamellar ichthyosis |
| X78CE | Non-erythrodermic lamellar ichthyosis |
| X78CF | Autosomal dominant lamellar ichthyosis |
| X78CG | Non-bullous ichthyosiform erythroderma |
| X3085 | Ichthyosis congenita with biliary atresia |
| X78CH | Bullous ichthyosis |
| X78CI | Bullous ichthyosiform erythroderma |
| X78CJ | Localised bullous ichthyosiform erythroderma |
| X78CK | Ichthyosis bullosa of Siemens |
| PH11. | Harlequin ichthyosis |
| X78CL | Ichthyosis hystrix |
| X78CM | Ichthyosis hystrix of Curth-Macklin |
| X78CN | Maleformatio ectodermalis generalisata of Bafverstedt |
| X78CO | Ichthyosis hystrix gravior of Rheydt |
| X78CP | Hystrix ichthyosis with deafness |
| X78CQ | Porcupine man |
| PH10. | Congenital ichthyosis, unspecified |
| PH1y. | Other specified ichthyosis congenita |
| XE1ML | Ichthyosis congenita NOS |
| Pyu90 | [X]Other congenital ichthyosis |
| XE1MK | Ichthyosiform erythroderma |
| X78C7 | Congenital ichthyosiform erythroderma |
| X507Q | Acquired ichthyosis |
| X501K | Keratitis ichthyosis and deafness syndrome |
| X50IM | Atypical ichthyosis vulgaris with hypogonadism |
| X78BT | Nethertons syndrome |
| SNOMED CT ID | Description |
| 111303009 | Ichthyosiform erythroderma |
| 111303003 | i intergration of year oder the |

| 12215009 | Recessive congenital ichthyosiform erythroderma |
|---|---|
| 13059002 | Ichthyosis congenita |
| 157017000 | Integument anomalies: [ichthyosis congenita] or [Dariers] or [keratosis follicularis] or [Meiges] or [Milroys] or [Mongolian spots] or [pseudoxanthoma elasticum] or [congenital NOS] |
| 19604005 | Triglyceride storage disease with ichthyosis |
| 201053002 | (Acquired ichthyosis) or (acquired keratoderma) or (hyperkeratosis NOS) |
| 201058006 | Acquired ichthyosis |
| 20512000 | Dominant congenital ichthyosiform erythroderma |
| 205547001 | Congenital ichthyosis, unspecified |
| 205548006 | Harlequin ichthyosis |
| 205549003 | Ichthyosiform erythroderma |
| 205550003 | Collodion baby |
| 205551004 | Ichthyosis vulgaris |
| 205552006 | X-linked recessive ichthyosis |
| 205553001 | Other specified ichthyosis congenita |
| 205555008 | Nethertons syndrome |
| 205556009 | (Congenital ichthyosiform erythroderma) or (alligator skin) or (ichthyosis congenita NOS) |
| 205974009 | [X]Other congenital ichthyosis |
| 2355008 | Dwarfism-ichthyosiform erythroderma-mental deficiency syndrome |
| 235916001 | Ichthyosis congenita with biliary atresia |
| 238627002 | Follicular ichthyosis |
| 238997007 | Drug-induced ichthyosiform reaction |
| 239057002 | Cutaneous syndrome with ichthyosis |
| 239058007 | Nethertons syndrome |
| 239059004 | Keratitis ichthyosis and deafness syndrome |
| 239060009 | Atypical ichthyosis vulgaris with hypogonadism |
| 239061008 | Keratosis pilaris with ichthyosis and deafness |
| 254127001 | Nethertons syndrome |
| 254128006 | Recessive congenital ichthyosiform erythroderma |
| 254156001 | Ichthyosis congenita NOS |
| 254157005 | Ichthyosis vulgaris |
| 254158000 | Autosomal dominant ichthyosis vulgaris |
| 254160003 | X-linked recessive ichthyosis |
| 254161004 | Erythrodermic lamellar ichthyosis |
| 254163001 | Non-erythrodermic lamellar ichthyosis |
| 254164007 | Autosomal dominant lamellar ichthyosis |
| 254165008 | Non-bullous ichthyosiform erythroderma |
| 254166009 | Bullous ichthyosis |
| 254167000 | Bullous ichthyosiform erythroderma |
| 254168005 | Localised bullous ichthyosiform erythroderma |
| 254169002 | Ichthyosis bullosa of Siemens |
| 254170001 | Ichthyosis hystrix of Curth-Macklin |
| 254171002 | Maleformatio ectodermalis generalisata of Bafverstedt |
| 254172009 | Ichthyosis hystrix gravior of Rheydt |
| 254173004 | Hystrix ichthyosis with deafness |
| 254174005 | Porcupine man |

| 255425009 | Ichthyosiform |
|---|---|
| 2625009 | Keratosis-ichthyosis-deafness syndrome |
| 267372009 | Congenital non bullous ichthyosiform erythroderma |
| 268245001 | Harlequin fetus |
| 268282005 | Ichthyosiform erythroderma |
| 268283000 | Ichthyosis congenita NOS |
| | Ichthyosis congenita |
| 268355000 | · |
| 312514006 | Nethertons syndrome |
| 34638006 | Lamellar ichthyosis AND trichorrhexis invaginata syndrome |
| 3944006 | X-linked ichthyosis |
| 396228006 | Ichthyosis - acquired |
| 400166009 | Ichthyosis - acquired |
| 402368008 | Ichthyosiform sarcoidosis (disorder) |
| 402770002 | Autosomal dominant ichthyosis (disorder) |
| 402771003 | X-linked recessive ichthyosis (disorder) |
| 402772005 | Autosomal recessive ichthyosis (disorder) |
| 403777006 | Lamellar ichthyosis (limited type) (disorder) |
| 403778001 | X-linked dominant ichthyosis (Happle) |
| 403779009 | Ichthyosis, cerebellar degeneration and hepatosplenomegaly (disorder) |
| 403780007 | Autosomal recessive keratitis-ichthyosis-deafness syndrome (disorder) |
| | Photosensitivity with ichthyosis, brittle hair, impaired intelligence, |
| 403781006 | decreased fertility and short stature syndrome |
| 403782004 | Ichthyosis follicularis with alopecia and photophobia (IFAP) (disorder) |
| 54336006 | Ichthyosis linearis circumflexa |
| 55846006 | Ichthyosis of eyelid |
| 67510007 | Ichthyosis hystrix |
| 68551007 | Limb reduction-ichthyosis syndrome |
| 699315005 | Neutral lipid storage disease without ichthyosis |
| 703504006 | Congenital reticular ichthyosiform erythroderma (disorder) |
| 716097001 | Ichthyosis cheek eyebrow syndrome (disorder) |
| 717041008 | Syndromic recessive X-linked ichthyosis (disorder) |
| 717183001 | Keratoderma hereditarium mutilans with ichthyosis syndrome (disorder) |
| 718631006 | Annular epidermolytic ichthyosis (disorder) |
| 720639008 | Coloboma, congenital heart disease, ichthyosiform dermatosis, intellectual disability ear anomaly syndrome (disorder) |
| 722225007 | Intellectual disability, enteropathy, deafness, peripheral neuropathy, |
| 722035007 | ichthyosis, keratoderma syndrome (disorder) |
| 722114007 | Osteosclerosis, ichthyosis, premature ovarian failure syndrome |
| 722385008 | Cerebral dysgenesis, neuropathy, ichthyosis, palmoplantar keratoderma syndrome (disorder) |
| 724277002 | Congenital ichthyosis with hypotrichosis syndrome (disorder) |
| | Neonatal sclerosing cholangitis, ichthyosis, hypotrichosis syndrome |
| 724278007 | (disorder) |
| 724837004 | Keratinopathic ichthyosis (disorder) |
| 72523005 | Sex-linked ichthyosis |
| 725588002 | Bathing suit ichthyosis (disorder) |
| 732950006 | Ichthyosis, oral and digital anomalies syndrome |
| 732952003 | Congenital cataract ichthyosis syndrome |
| 733028000 | Multiple sclerosis, ichthyosis, factor VIII deficiency syndrome |

| 733097003 | Ichthyosis, intellectual disability, dwarfism, renal impairment syndrome (disorder) |
|---|---|
| 763401009 | Congenital ichthyosis type 4 |
| 763404001 | Ichthyosis, alopecia, eclabion, ectropion, intellectual disability syndrome |
| 763768001 | Autosomal recessive exfoliative ichthyosis (disorder) |
| 763775000 | Keratosis linearis, ichthyosis congenita, sclerosing keratoderma syndrome (disorder) |
| 765471005 | X-linked intellectual disability, hypogonadism, ichthyosis, obesity, short stature syndrome |
| 782957005 | Ichthyosis |
| 783551005 | Ichthyosis, short stature, brachydactyly, microspherophakia syndrome |
| 8691004 | Ichthyosis - acquired |
| 95334005 | Senile ichthyosis |

Diagnosis codes which will be used to identify VTE events.

| Pulmonary Embolism | |
|---|---|
| Read V2 Code | Code description |
| G401. | Pulmonary embolism |
| G4010 | Post operative pulmonary embolus |
| G4011 | Recurrent pulmonary embolism |
| L43 | Obstetric pulmonary embolism |
| L432. | Obstetric blood-clot pulmonary embolism |
| L4320 | Obstetric blood-clot pulmonary embolism unspecified |
| L4321 | Obstetric blood-clot pulmonary embolism - delivered |
| L4322 | Obstetric blood-clot pulmonary embolism - delivered with postnatal complication |
| L4323 | Obstetric blood-clot pulmonary embolism with antenatal complication |
| L4324 | Obstetric blood-clot pulmonary embolism with postnatal complication |
| L432z | Obstetric blood-clot pulmonary embolism NOS |
| L43y. | Other obstetric pulmonary embolism |
| L43y0 | Other obstetric pulmonary embolism unspecified |
| L43y1 | Other obstetric pulmonary embolism - delivered |
| L43y2 | Other obstetric pulmonary embolism - delivered with postnatal complication |
| L43y3 | Other obstetric pulmonary embolism with antenatal complication |
| L43y4 | Other obstetric pulmonary embolism with postnatal complication |
| L43yz | Other obstetric pulmonary embolism NOS |
| L43z. | Obstetric pulmonary embolism NOS |
| L43z0 | Obstetric pulmonary embolism NOS, unspecified |
| L43z1 | Obstetric pulmonary embolism NOS - delivered |
| L43z2 | Obstetric pulmonary embolism NOS - delivered with postnatal complication |
| L43z3 | Obstetric pulmonary embolism NOS with antenatal complication |
| L43z4 | Obstetric pulmonary embolism NOS with postnatal complication |
| L43zz | Obstetric pulmonary embolism NOS |
| L0964 | Pulmonary embolism following abortive pregnancy |
| Read CTV3 Code | Description |
| XE0Um | Pulmonary embolus |
| XaOYV | Recurrent pulmonary embolism |
| X202x | Pulmonary thromboembolism |
| X202y | Acute massive pulmonary embolism |
| X202z | Subacute massive pulmonary embolism |
| G4010 | Postoperative pulmonary embolus |
| L43 | Obstetric pulmonary embolism |
| L432. | Obstetric blood-clot pulmonary embolism |
| L4320 | Obstetric blood-clot pulmonary embolism unspecified |
| L4321 | Obstetric blood-clot pulmonary embolism - delivered |
| L4322 | Obstetric blood-clot pulmonary embolism - delivered with postnatal complication |
| L4323 | Obstetric blood-clot pulmonary embolism with antenatal complication |

| L4324 | Obstetric blood-clot pulmonary embolism with postnatal complication |
|---|---|
| L432z | Obstetric blood-clot pulmonary embolism NOS |
| L43z. | Obstetric pulmonary embolism NOS |
| L43z0 | Obstetric pulmonary embolism NOS, unspecified |
| L43z1 | Obstetric pulmonary embolism NOS - delivered |
| | Obstetric pulmonary embolism NOS - delivered with postnatal |
| L43z2 | complication |
| L43z3 | Obstetric pulmonary embolism NOS with antenatal complication |
| L43z4 | Obstetric pulmonary embolism NOS with postnatal complication |
| XE0xN | Other obstetric pulmonary embolism |
| L43y0 | Other obstetric pulmonary embolism unspecified |
| L43y1 | Other obstetric pulmonary embolism - delivered |
| L43y2 | Other obstetric pulmonary embolism - delivered with postnatal complication |
| L43y3 | Other obstetric pulmonary embolism with antenatal complication |
| L43y4 | Other obstetric pulmonary embolism with postnatal complication |
| L43yz | Other obstetric pulmonary embolism NOS |
| X012b | Operation for pulmonary embolism |
| X012c | Embolectomy of pulmonary artery |
| 7A0A1 | Percutaneous embolectomy of pulmonary artery |
| 7A093 | Open pulmonary embolectomy |
| X012d | Transluminal fragmentation of pulmonary embolus |
| XaBMd | [V] Personal history of pulmonary embolism |
| L0964 | |
| 14AC. | Pulmonary embolism following abortive pregnancy H/O: pulmonary embolus |
| SNOMED CT ID | Description |
| 155326007 | (Pulmonary embolism) or (pulmonary infarct) (disorder) |
| 308159008 | [V] Personal history of pulmonary embolism |
| 315761003 | [V] Personal history of pulmonary embolism |
| 50206009 | Abortion with pulmonary embolism |
| 706870000 | Acute pulmonary embolism |
| 17263003 | Amniotic fluid pulmonary embolism |
| 200294005 | Amniotic fluid pulmonary embolism - delivered (disorder) Amniotic fluid pulmonary embolism - delivered with postnatal |
| 200295006 | complication (disorder) |
| 200298008 | Amniotic fluid pulmonary embolism NOS (disorder) |
| 200293004 | Amniotic fluid pulmonary embolism unspecified (disorder) |
| 200296007 | Amniotic fluid pulmonary embolism with antenatal complication (disorder) |
| 200297003 | Amniotic fluid pulmonary embolism with postnatal complication (disorder) |
| 233936003 | AMPE - Acute massive pulmonary embolism |
| 133971000119108 | Chronic pulmonary embolism |
| | Failed attempted abortion with pulmonary embolism |
| 58123006 | Failed attempted abortion with pulmonary embolism |
| | Failed attempted abortion with pulmonary embolism Family history of pulmonary embolism (situation) |
| 58123006 | |
| 58123006<br>430801003 | Family history of pulmonary embolism (situation) |
| 58123006<br>430801003<br>10761511000119101 | Family history of pulmonary embolism (situation) History of pulmonary embolism on long-term anticoagulation therapy |

| 200288002 | Obstetric air pulmonary embolism - delivered (disorder) |
|---|---|
| 200289005 | Obstetric air pulmonary embolism - delivered with postnatal complication (disorder) |
| 200286003 | Obstetric air pulmonary embolism (disorder) |
| 200292009 | Obstetric air pulmonary embolism NOS (disorder) |
| 200287007 | Obstetric air pulmonary embolism unspecified (disorder) |
| 200290001 | Obstetric air pulmonary embolism with antenatal complication (disorder) |
| 200291002 | Obstetric air pulmonary embolism with postnatal complication (disorder) |
| 200301007 | Obstetric blood-clot pulmonary embolism - delivered (disorder) |
| 200302000 | Obstetric blood-clot pulmonary embolism - delivered with postnatal complication |
| 200299000 | Obstetric blood-clot pulmonary embolism (disorder) |
| 200305003 | Obstetric blood-clot pulmonary embolism NOS |
| 200300008 | Obstetric blood-clot pulmonary embolism unspecified (disorder) |
| 200303005 | Obstetric blood-clot pulmonary embolism with antenatal complication |
| 200304004 | Obstetric blood-clot pulmonary embolism with postnatal complication |
| 237341004 | Obstetric pulmonary embolism |
| 156273009 | Obstetric pulmonary embolism (disorder) |
| 200320009 | Obstetric pulmonary embolism NOS |
| 200326003 | Obstetric pulmonary embolism NOS |
| 200322001 | Obstetric pulmonary embolism NOS - delivered |
| 200323006 | Obstetric pulmonary embolism NOS - delivered with postnatal complication |
| 200324000 | Obstetric pulmonary embolism NOS with antenatal complication |
| 200325004 | Obstetric pulmonary embolism NOS with postnatal complication |
| 200321008 | Obstetric pulmonary embolism NOS, unspecified |
| 267284008 | Obstetric pyaemic and septic pulmonary embolism |
| 200308001 | Obstetric pyaemic and septic pulmonary embolism - delivered |
| 200312007 | Obstetric pyaemic and septic pulmonary embolism NOS |
| 200310004 | Obstetric pyaemic and septic pulmonary embolism with antenatal complication |
| 200306002 | Obstetric pyemic and septic pulmonary embolism |
| 200309009 | Obstetric pyemic and septic pulmonary embolism - delivered with postnatal complication |
| 200307006 | Obstetric pyemic and septic pulmonary embolism unspecified |
| 200244000 | Obstetric pyemic and septic pulmonary embolism with postnatal |
| 200311000 | complication |
| 50286006 | Obstetrical pulmonary embolism |
| 233217004 | Operation for pulmonary embolism |
| 200313002 | Other obstetric pulmonary embolism |
| 267285009 | Other obstetric pulmonary embolism |
| 200315009 | Other obstetric pulmonary embolism - delivered (disorder) Other obstetric pulmonary embolism - delivered with postnatal |
| 200316005 | complication (disorder) |
| 200319003 | Other obstetric pulmonary embolism NOS |
| 200314008 | Other obstetric pulmonary embolism unspecified (disorder) |
| 200317001 | Other obstetric pulmonary embolism with antenatal complication |
| 200318006 | Other obstetric pulmonary embolism with postnatal complication |

| 45015000 | Other obstetrical pulmonary embolism, NEC |
|---|---|
| 200284000 | Puerperal pulmonary embolism |
| 194882001 | Pulmonary embolism |
| 266292008 | Pulmonary embolism Pulmonary embolism |
| 59282003 | Pulmonary embolism |
| 39202003 | Pulmonary embolism as current complication following acute |
| 723859005 | myocardial infarction (disorder) |
| 860680001 | Pulmonary embolism due to and following ectopic pregnancy |
| 860681002 | Pulmonary embolism due to and following molar pregnancy (disorder) |
| 198855003 | Pulmonary embolism following abortive pregnancy |
| 663008 | Pulmonary embolism following molar AND/OR ectopic pregnancy |
| 10759311000119104 | Pulmonary embolism in childbirth (disorder) |
| 713078005 | Pulmonary embolism on long-term anticoagulation therapy (disorder) |
| 1001000119102 | Pulmonary embolism with infarction |
| 438773007 | Recurrent pulmonary embolism (disorder) |
| 441557008 | Septic pulmonary embolism |
| 82153002 | Spontaneous abortion with pulmonary embolism |
| 233937007 | Subacute massive pulmonary embolism |
| 417113001 | Suspected pulmonary embolism (context-dependent category) |
| 609480009 | Termination of pregnancy complicated by pulmonary embolism |
| 82153002 | Miscarriage with pulmonary embolism (disorder) |
| 860681002 | Pulmonary embolism due to and following molar pregnancy (disorder) |
| Deep Vein Thrombosis | |
| Read V2 Code | Code description |
| G801. | Deep vein thrombosis |
| G8010 | Phlebitis of the femoral vein |
| G8011 | Phlebitis of the popliteal vein |
| G8012 | Phlebitis of the anterior tibial vein |
| i | |
| G8013 | Phlebitis of the dorsalis pedis vein |
| G8013<br>G8014 | Phlebitis of the dorsalis pedis vein Phlebitis of the posterior tibial vein |
| | · |
| G8014 | Phlebitis of the posterior tibial vein |
| G8014<br>G8015 | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified |
| G8014<br>G8015<br>G8016 | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the femoral vein |
| G8014<br>G8015<br>G8016<br>G8017 | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the femoral vein Thrombophlebitis of the popliteal vein |
| G8014<br>G8015<br>G8016<br>G8017<br>G8018 | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the femoral vein Thrombophlebitis of the popliteal vein Thrombophlebitis of the anterior tibial vein |
| G8014<br>G8015<br>G8016<br>G8017<br>G8018<br>G8019 | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the femoral vein Thrombophlebitis of the popliteal vein Thrombophlebitis of the anterior tibial vein Thrombophlebitis of the dorsalis pedis vein |
| G8014<br>G8015<br>G8016<br>G8017<br>G8018<br>G8019<br>G801A | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the femoral vein Thrombophlebitis of the popliteal vein Thrombophlebitis of the anterior tibial vein Thrombophlebitis of the dorsalis pedis vein Thrombophlebitis of the posterior tibial vein |
| G8014<br>G8015<br>G8016<br>G8017<br>G8018<br>G8019<br>G801A<br>G801B | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the femoral vein Thrombophlebitis of the popliteal vein Thrombophlebitis of the anterior tibial vein Thrombophlebitis of the dorsalis pedis vein Thrombophlebitis of the posterior tibial vein Deep vein thrombophlebitis of the leg unspecified |
| G8014<br>G8015<br>G8016<br>G8017<br>G8018<br>G8019<br>G801A<br>G801B<br>G801C | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the femoral vein Thrombophlebitis of the popliteal vein Thrombophlebitis of the anterior tibial vein Thrombophlebitis of the dorsalis pedis vein Thrombophlebitis of the posterior tibial vein Deep vein thrombophlebitis of the leg unspecified Deep vein thrombosis of leg related to air travel |
| G8014 G8015 G8016 G8017 G8018 G8019 G801A G801B G801C G801D | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the femoral vein Thrombophlebitis of the popliteal vein Thrombophlebitis of the anterior tibial vein Thrombophlebitis of the dorsalis pedis vein Thrombophlebitis of the posterior tibial vein Deep vein thrombophlebitis of the leg unspecified Deep vein thrombosis of leg related to air travel Deep vein thrombosis of lower limb |
| G8014 G8015 G8016 G8017 G8018 G8019 G801A G801B G801C G801D G801E | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the popliteal vein Thrombophlebitis of the anterior tibial vein Thrombophlebitis of the dorsalis pedis vein Thrombophlebitis of the posterior tibial vein Deep vein thrombophlebitis of the leg unspecified Deep vein thrombosis of leg related to air travel Deep vein thrombosis of lower limb Deep vein thrombosis of leg related to intravenous drug use |
| G8014 G8015 G8016 G8017 G8018 G8019 G801A G801B G801C G801D G801E G801F | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the femoral vein Thrombophlebitis of the popliteal vein Thrombophlebitis of the anterior tibial vein Thrombophlebitis of the dorsalis pedis vein Thrombophlebitis of the posterior tibial vein Deep vein thrombophlebitis of the leg unspecified Deep vein thrombosis of leg related to air travel Deep vein thrombosis of lower limb Deep vein thrombosis of leg related to intravenous drug use Deep vein thrombosis of peroneal vein |
| G8014 G8015 G8016 G8017 G8018 G8019 G801A G801B G801C G801D G801E G801F G801G | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the popliteal vein Thrombophlebitis of the anterior tibial vein Thrombophlebitis of the dorsalis pedis vein Thrombophlebitis of the posterior tibial vein Deep vein thrombophlebitis of the leg unspecified Deep vein thrombosis of leg related to air travel Deep vein thrombosis of lower limb Deep vein thrombosis of leg related to intravenous drug use Deep vein thrombosis of peroneal vein Recurrent deep vein thrombosis |
| G8014 G8015 G8016 G8017 G8018 G8019 G801A G801B G801C G801D G801E G801F G801G G801H | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the femoral vein Thrombophlebitis of the popliteal vein Thrombophlebitis of the anterior tibial vein Thrombophlebitis of the dorsalis pedis vein Thrombophlebitis of the posterior tibial vein Deep vein thrombophlebitis of the leg unspecified Deep vein thrombosis of leg related to air travel Deep vein thrombosis of lower limb Deep vein thrombosis of leg related to intravenous drug use Deep vein thrombosis of peroneal vein Recurrent deep vein thrombosis Unprovoked deep vein thrombosis |
| G8014 G8015 G8016 G8017 G8018 G8019 G801A G801B G801C G801D G801E G801F G801G G801H | Phlebitis of the posterior tibial vein Deep vein phlebitis of the leg unspecified Thrombophlebitis of the popliteal vein Thrombophlebitis of the anterior tibial vein Thrombophlebitis of the dorsalis pedis vein Thrombophlebitis of the posterior tibial vein Deep vein thrombophlebitis of the leg unspecified Deep vein thrombosis of leg related to air travel Deep vein thrombosis of lower limb Deep vein thrombosis of leg related to intravenous drug use Deep vein thrombosis of peroneal vein Recurrent deep vein thrombosis Unprovoked deep vein thrombosis Provoked deep vein thrombosis |

| L414. | Postnatal deep vein thrombosis |
|---|---|
| L4140 | Postnatal deep vein thrombosis unspecified |
| L4141 | Postnatal deep vein thrombosis - delivered with postnatal complication |
| L4142 | Postnatal deep vein thrombosis with postnatal complication |
| L414z | Postnatal deep vein thrombosis NOS |
| L413. | Antenatal deep vein thrombosis |
| L4130 | Antenatal deep vein thrombosis unspecified |
| L4131 | Antenatal deep vein thrombosis - delivered |
| L4132 | Antenatal deep vein thrombosis with antenatal complication |
| L413z | Antenatal deep vein thrombosis NOS |
| 14A81 | H/O: Deep Vein Thrombosis |
| ZV128 | [V] Personal history DVT - deep vein thrombosis |
| G8020 | Thrombosis of vein of leg |
| Read CTV3 Code | Description |
| Xa9Bs | Deep vein thrombosis |
| X205n | lleofemoral deep vein thrombosis |
| X205m | Lower venous segment thrombosis |
| XaQIV | Deep venous thrombosis of peroneal vein |
| X76Lg | Phlegmasia alba dolens |
| Xa1aj | Phlegmasia alba dolens - obstetric |
| X76Lh | Phlegmasia caerula dolens |
| SP122 | Postoperative deep vein thrombosis |
| L413. | Antenatal deep vein thrombosis |
| L4130 | Antenatal deep vein thrombosis unspecified |
| L4131 | Antenatal deep vein thrombosis - delivered |
| L4132 | Antenatal deep vein thrombosis with antenatal complication |
| L413z | Antenatal deep vein thrombosis NOS |
| XE0xL | Postnatal deep vein thrombosis |
| L4140 | Postnatal deep vein thrombosis unspecified |
| L4141 | Postnatal deep vein thrombosis - delivered with postnatal complication |
| L4142 | Postnatal deep vein thrombosis - delivered with postnatal complication |
| L414z | Postnatal deep vein thrombosis NOS |
| XaJxo | Deep vein thrombosis of leg related to intravenous drug use |
| Xallo | Deep vein thrombosis of leg related to intravellous drug use Deep vein thrombosis of leg related to air travel |
| Xacve | Provoked deep vein thrombosis |
| Xacve | Unprovoked deep vein thrombosis |
| XaZ43 | Recurrent deep vein thrombosis |
| XaCOs | Thrombosis of vein of lower limb |
| | [V] Personal history DVT - deep vein thrombosis |
| XaBMc | |
| 14A81 | H/O: Deep Vein Thrombosis |
| XaaBG | On deep vein thrombosis care pathway |
| XEOVY | Deep vein phlebitis and thrombophlebitis of the leg |
| G801z | Deep vein phlebitis and thrombophlebitis of the leg NOS |
| X205e | Deep thrombophlebitis |
| Xa205l | High venous segment venous thrombosis |
| G8016 | Thrombophlebitis of femoral vein |
| G8017 | Thrombophlebitis of popliteal vein |

| G801B | Thrombophebitis of the leg unspecified |
|---|---|
| G802. | Phlebitis and thrombophlebitis of leg NOS |
| Gyu80 | [X] Phlebitis and thrombophlebitis/oth deep vessls/low extremites |
| SNOMED CT ID | Description |
| 195403006 | (Deep vein phlebitis and thrombophlebitis of the leg) or (deep vein thrombosis) |
| 315760002 | [V] Personal history deep vein thrombosis |
| 285381000119104 | Acute deep vein thrombosis of bilateral femoral veins |
| 293491000119107 | Acute deep vein thrombosis of left iliac vein |
| 15711401000119105 | Acute deep vein thrombosis of left lower limb following procedure |
| 651000119108 | Acute deep vein thrombosis of lower limb (disorder) |
| 293481000119109 | Acute deep vein thrombosis of right iliac vein |
| 15708401000119100 | Acute deep vein thrombosis of right lower limb following procedure |
| 15708201000119101 | Acute deep vein thrombosis of right upper limb following procedure |
| 132251000119101 | Acute deep venous thrombosis of popliteal vein (disorder) |
| 132271000119105 | Acute deep venous thrombosis of thigh (disorder) |
| 285381000119104 | Acute deep vein thrombosis of bilateral femoral veins (disorder) |
| | Acute deep venous thrombosis of lower extremity as complication of |
| 136781000119101 | procedure (disorder) |
| 132261000119104 | Acute deep venous thrombosis of tibial vein (disorder) |
| 134961000119104 | Acute deep venous thrombosis of axillary vein (disorder) |
| 156268003 | Antenatal deep vein thrombosis |
| 200232006 | Antenatal deep vein thrombosis - delivered |
| 200234007 | Antenatal deep vein thrombosis NOS |
| 200231004 | Antenatal deep vein thrombosis unspecified |
| 200233001 | Antenatal deep vein thrombosis with antenatal complication |
| 49956009 | Antepartum deep vein thrombosis |
| 225999004 | At risk of deep vein thrombosis |
| 293461000119100 | Chronic deep vein thrombosis of left iliac vein (disorder) |
| 709687000 | Chronic deep vein thrombosis of pelvic vein |
| 293451000119102 | Chronic deep vein thrombosis of right iliac vein |
| 132131000119102 | Chronic deep venous thrombosis of calf (disorder) |
| 132191000119103 | Chronic deep venous thrombosis of femoral vein (disorder) |
| 132201000119100 | Chronic deep venous thrombosis of iliofemoral vein (disorder) |
| 503421000000105 | Deep vein thrombosis enhanced services administration stage 1 service level (finding) |
| 132141000119106 | Chronic deep venous thrombosis of lower extremity (disorder) |
| 132091000119104 | Chronic deep venous thrombosis of lower limb due to coronary artery bypass grafting (disorder) |
| 132151000119108 | Chronic deep venous thrombosis of popliteal vein (disorder) |
| 132171000119104 | Chronic deep venous thrombosis of thigh (disorder) |
| 132221000119109 | Chronic deep venous thrombosis of upper extremity (disorder) |
| 136751000119108 | Chronic deep venous thrombosis of upper extremity as complication of procedure (disorder) |
| 503451000000100 | Deep vein thrombosis enhanced services administration stage 2 service level (finding) |
| 503481000000106 | Deep vein thrombosis enhanced services administration stage 3 service level (finding) |
| 132551000119104 | Chronic thrombosis of subclavian vein (disorder) |
| 16750002 | Deep thrombophlebitis |

| 444325005 | Deep vein thrombosis of bilateral lower extremities (disorder) |
|---|---|
| 134399007 | Deep vein thrombosis of leg related to air travel |
| 366830006 | Deep vein thrombosis of leg related to air travel |
| 366911007 | Deep vein thrombosis of leg related to air travel |
| 413956008 | Deep vein thrombosis of leg related to intravenous drug use (disorder) |
| 860699005 | Deep vein thrombosis of lower extremity due to intravenous drug use |
| 366912000 | Deep vein thrombosis of lower limb |
| 17920008 | Deep vein thrombosis of portal vein |
| 14534009 | Deep vein thrombosis of splenic vein |
| 401186003 | Deep vein thrombosis screening |
| 155454004 | Deep vein thrombosis-non obst. |
| 266328001 | Deep vein thrombosis-non obst. |
| 267361004 | Deep vein thrombosis-obstetric |
| 128053003 | DVT |
| 128057002 | DVT - Deep vein thrombosis of lower limb |
| 404223003 | DVT - Deep vein thrombosis of lower limb |
| 200235008 | DVT: [postnatal] or [obstetric phlegmasia alba dolens] |
| | Deep venous thrombosis of tibial vein (disorder) |
| 438785004 | . , |
| 132161000119105 | Chronic deep venous thrombosis of tibial vein (disorder) |
| 703277001 | Deep venous thrombosis of femoropopliteal vein (disorder) |
| 427775006 | Deep venous thrombosis of profunda femoris vein (disorder) |
| 161508001 | History of deep vein thrombosis |
| 141911000119100 | History of recurrent deep vein thrombosis |
| 234044007 | Ileofemoral deep vein thrombosis |
| 156264001 | Obstetric venous problems (& [deep vein thrombosis] or [varicose vein]) (disorder) |
| 156269006 | Postnatal deep vein thrombosis |
| 200237000 | Postnatal deep vein thrombosis - delivered with postnatal complication |
| 200239002 | Postnatal deep vein thrombosis NOS |
| 200236009 | Postnatal deep vein thrombosis unspecified |
| 200238005 | Postnatal deep vein thrombosis with postnatal complication |
| 213220000 | Postoperative deep vein thrombosis |
| 56272000 | Postpartum deep vein thrombosis |
| 439993001 | Prevention of deep vein thrombosis (regime/therapy) |
| 710167004 | Recurrent deep vein thrombosis (disorder) |
| 431883007 | Referral to deep vein thrombosis clinic (procedure) |
| 432805000 | Suspected deep vein thrombosis (situation) |
| 978441000000108 | Provoked deep vein thrombosis (disorder) |
| 978421000000101 | Unprovoked deep vein thrombosis (disorder) |
| 869721000000104 | Deep vein thrombosis care pathway (regime/therapy) |
| 128055005 | Deep venous thrombosis of pelvic vein (disorder) |
| 443210003 | Deep venous thrombosis of peroneal vein (disorder) |
| 141911000119100 | History of recurrent deep vein thrombosis (situation) |
| | Acute deep vein thrombosis of left lower limb following coronary artery |
| 15708361000119109 | bypass graft (disorder) |
| 45700244000446464 | Acute deep vein thrombosis of right lower limb following coronary |
| 15708241000119104 | artery bypass graft (disorder) |
| 429098002 | Thromboembolism of vein (disorder) |

Below is a list of the variables to be extracted and utilised for the study

| Variable | Role | Data source(s) | Operational |
|---|---|---|---|
| | | | definition |
| Atopic Dermatitis | Case definition | OPCRD | As defined using the |
| | | | codes listed in |
| | | | Appendix 1 |
| Atopic Dermatitis | Case definition | OPCRD | As defined using the |
| severity | | | codes listed in |
| | | | Appendix 1 and the |
| | | | approach described in |
| | | | section 3.4. |
| Atopic Dermatitis | Case definition | OPCRD | As defined using the |
| exclusion conditions | | | codes listed in |
| | | | Appendix 2 |
| Pulmonary embolism | Study outcome | OPCRD | As defined using the |
| (PE) | | | codes listed in |
| | | | Appendix 3 |
| Deep vein thrombosis | Study outcome | OPCRD | As defined using the |
| (DVT) | | | codes listed in |
| | | | Appendix 3 |
| Age | Baseline characteristic, | OPCRD | Defined as age at the |
| | predictor variable | | start of follow up |
| Gender | Baseline characteristic, | OPCRD | Primary care recorded |
| | predictor variable | | patient gender |
| Socioeconomic status | Baseline characteristic, | OPCRD | Defined using patient |
| (SES) | predictor variable | | index of multiple |
| | | | deprivation quintile |
| Ethnicity | Baseline characteristic, | OPCRD | Defined using office of |
| | predictor variable | | national statistics |
| | | | census categories using |
| | | | clinically coded |
| | | | ethnicity data |
| Smoking status | Baseline characteristic, | OPCRD | Using most recent |
| | predictor variable | | clinically recorded |
| | | | smoking status |
| | | | information |
| Alcohol use | Baseline characteristic, | OPCRD | Using most recent |
| | predictor variable | | clinically recorded |

| | | 1 | alcohol use status |
|---|---|---|---|
| | | | information |
| Body mass index (BMI) | Baseline characteristic, | OPCRD | Defined using most |
| | predictor variable | | recent clinically |
| | | | recorded BMI |
| | | | information |
| Death | Censoring event | OPCRD | Identified from coding |
| | | | in the clinical record |
| Deregistration from GP | Censoring event | OPCRD | Identified from coding |
| | | | in the clinical record |
| Atrial fibrillation | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Angina | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Myocardial infarction | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Congestive heart failure | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Stroke | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Diabetes type | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Hyperlipidaemia | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| | Baseline characteristic, | OPCRD | Identified using clinical |
| Hypertension | predictor variable | | codes for the condition |
| Cl . 1 . 1 . 1 | Baseline characteristic, | OPCRD | Identified using clinical |
| Chronic kidney disease | predictor variable | | codes for the condition |
| stages 3-5 | | | and lab test results |
| Chronic obstructive | Baseline characteristic, | OPCRD | Identified using clinical |
| pulmonary disease, | predictor variable | | codes for the condition |
| Asthma | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Chronic liver disease | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Dementia | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Immunotherapy use | Potential predictor | OPCRD | Identified using |
| | variable | | prescription records for |
| | | | immunotherapy |
| | | 1 | |

| Phototherapy | Potential predictor | OPCRD | Identified using |
|--------------|---------------------|-------|------------------------|
| treatment | variable | | prescription records |
| | | | and clinical codes for |
| | | | phototherapy |